CLINICAL TRIAL: NCT00908037
Title: A Three Part, Staggered Cohort, Open-label and Double Blind, Randomized, Placebo Controlled Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of Eltrombopag, a Thrombopoietin Receptor Agonist, in Previously Treated Pediatric Patients With Chronic ITP.
Brief Title: Efficacy and Safety Study of Eltrombopag in Pediatric Patients With Thrombocytopenia From Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Acronym: PETIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108062
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2015-03

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: idiopathic thrombocytopenic purpura; thrombocytopenia; pharmacodynamics; ITP; eltrombopag; pharmacokinetics; chronic ITP; pediatrics
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eltrombopag plus standard of care (Experimental): eltrombopag
  Interventions: Drug: eltrombopag
- placebo plus standard of care (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eltrombopag — thrombopoietin receptor agonist
  Arms: eltrombopag plus standard of care
Drug: Placebo — placebo for comparison
  Arms: placebo plus standard of care

SUMMARY:
Phase II, multi-center, 3 part, staggered cohort, open-label and double blind, randomized, placebo controlled study involving 3 age-determined cohorts (Cohort 1: between 12 and 17 years old; Cohort 2: between 6 and 11 years old; Cohort 3: between 1 and 5 years old). Daily dosing with eltrombopag will begin with 5 patients in the oldest age cohort in an open label fashion, and a review of safety, pharmacokinetic and platelet count data will be performed regularly. If no safety concerns are identified after 12 weeks, 18 additional patients will be randomised to placebo or eltrombopag (2:1 randomisation). After 7 weeks of randomized treatment, all patients will receive eltrombopag in an open label fashion. The total duration of treatment with eltrombopag will be 24 weeks. If at the time of the aforementioned 12 week review of the first 5 patients no safety issues are identified, dosing will begin in the next lower age cohort with an initial group of 5 patients. The same procedure will be followed in terms of safety review and subsequent enrolment and randomisation of the additional patients. Initiation of the younger age cohort will take place once data from the previous has been evaluated. Doses will be adjusted according to platelet counts and tolerability. The study will include a review of the safety data by a Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 1 year and <18 years of age at Day 1.
* Written informed consent from subject's guardian and accompanying informed assent from subject (for children over 6 years old).
* Confirmed diagnosis of chronic ITP, according to the American Society of Hematology / British Committee for Standards in Haematology (ASH/BCSH) guidelines [George, 1996; BCSH, 2003]. In addition, a peripheral blood smear or bone marrow examination should support the diagnosis of ITP with no evidence of other causes of thrombocytopenia.
* Subjects who are refractory or have relapsed after at least one prior ITP therapy or are not eligible, for a medical reason, for other treatments.
* Day 1 (or within 48 hours prior) platelet count <30 Gi/L.
* Previous therapy for ITP with immunoglobulins (IVIg and anti-D) must have been completed at least 2 weeks prior to Day 1 or have been clearly ineffective.
* Subjects treated with concomitant ITP medication (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for at least 4 weeks prior to Day 1.
* Previous treatment for ITP with splenectomy, rituximab and cyclophosphamide must have been completed at least 4 weeks prior to Day 1 or have clearly been ineffective.
* Subjects must have prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) within 80 to 120% of the normal range.
* Subjects must have a complete blood count (CBC) not suggestive of another hematological disorder.
* The following clinical chemistries for the subjects MUST NOT exceed the upper limit of normal (ULN) reference range by more than 20%: creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and alkaline phosphatase. In addition, total albumin must not be below the lower limit of normal (LLN) by more than 10%.
* For subjects of child-bearing potential (after menarche): subject must not be sexually active or is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must use one of the following highly effective methods of contraception (i.e., Pearl Index <1.0%) from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:
* Complete abstinence from intercourse;
* Intrauterine device (IUD);
* Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide);
* Systemic contraceptives (combined or progesterone only).

Exclusion Criteria:

* Any clinically relevant abnormality, other than ITP, identified on the screening examination or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another primary diagnosis (e.g. thrombocytopenia is secondary to another disease).
* Concurrent or past malignant disease, including myeloproliferative disorder.
* Subjects who are not suitable for continuation of their current therapy for at least 7 additional additional weeks.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Day 1.
* History of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* Diagnosis of secondary immune thrombocytopenia, including those with laboratory or clinical evidence of HIV infection, anti-phospholipid antibody syndrome, chronic hepatitis B infection, hepatitis C virus infection, or any evidence of active hepatitis at the time of subject screening.
* Subject with Evans syndrome (autoimmune thrombocytopenia and autoimmune hemolysis).
* Subjects with known inherited thrombocytopenia (e.g. MYH-9 disorders)
* Subjects treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for >3 consecutive days within 2 weeks of Day 1.
* Subjects who have previously received eltrombopag or any other thrombopoietin receptor agonist.
* For female subjects who have reached menarche status, an inability or unwillingness to provide a blood or urine specimen for pregnancy testing.
* Female subjects who are pregnant or lactating.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2009-09-30; Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (17):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (2):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Paris
- GSK Investigational Site, Rotterdam, Netherlands
- Spain (3):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- United Kingdom (5):
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Southampton

REFERENCES:
- [Derived] Grainger JD, Blanchette VS, Grotzinger KM, Roy A, Bussel JB. Health-related quality of life in children with chronic immune thrombocytopenia treated with eltrombopag in the PETIT study. Br J Haematol. 2019 Apr;185(1):102-106. doi: 10.1111/bjh.15732. Epub 2018 Dec 27. PMID 30592022
- [Derived] Wire MB, Li X, Zhang J, Sallas W, Aslanis V, Ouatas T. Modeling and Simulation Support Eltrombopag Dosing in Pediatric Patients With Immune Thrombocytopenia. Clin Pharmacol Ther. 2018 Dec;104(6):1199-1207. doi: 10.1002/cpt.1066. Epub 2018 Apr 17. PMID 29536526
- [Derived] Bussel JB, de Miguel PG, Despotovic JM, Grainger JD, Sevilla J, Blanchette VS, Krishnamurti L, Connor P, David M, Boayue KB, Matthews DC, Lambert MP, Marcello LM, Iyengar M, Chan GW, Chagin KD, Theodore D, Bailey CK, Bakshi KK. Eltrombopag for the treatment of children with persistent and chronic immune thrombocytopenia (PETIT): a randomised, multicentre, placebo-controlled study. Lancet Haematol. 2015 Aug;2(8):e315-25. doi: 10.1016/S2352-3026(15)00114-3. Epub 2015 Jul 28. PMID 26688484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants (par.) meeting eligibility criteria were enrolled into 3 cohorts depending upon age. Cohort 1 enrolled participants who were between 12 and 17 years old, Cohort 2 enrolled participants who were between 6 and 11 years old, and Cohort 3 enrolled participants who were between 1 and 5 years old.
Pre-assignment Details: 15 par. were randomized to a 24-Week (Wk) Open-Label (OL) eltrombopag Dose-Finding period (pd) (Part 1) then did not continue. 67 par. were randomized to a 7-Wk Double-Blind placebo-controlled pd (Part 2), followed by a 24-Wk OL eltrombopag-only pd (Part 2/3) and a 4-Wk Follow-Up pd.
Groups:
- Part 1 (Dose-Finding Period) Cohort 1: Participants aged between 12 and 17 years received a 24-week Open-Label treatment of eltrombopag administered as a tablet. The starting dose of eltrombopag was 25 milligrams (mg), once daily (QD). The participants of East Asian ancestry began at 12.5 mg QD. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 1 (Dose-Finding Period) Cohort 2: Participants aged between 6 and 11 years received a 24-week Open-Label treatment of eltrombopag administered as a tablet. The starting dose of eltrombopag was based on the body weight. Participants with a weight of <27 kilograms (kg) received 12.5 mg QD (approximately 0.5 - 0.7 mg/kg QD) and participants with a weight of >=27 kg received 25 mg QD (approximately 0.5 - 0.8 mg/kg QD). The maximum dose allowed was 2 mg/kg and could not exceed 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 1 (Dose-Finding Period) Cohort 3: Participants aged between 1 and 5 years received a 24-week Open-Label treatment of eltrombopag administered as a dry powder for oral suspension. The starting dose of eltrombopag was 0.7 mg/kg QD. Participants of East Asian ancestry began at 0.5 mg/kg/day. The maximum dose allowed was 2 mg/kg, and could not exceed 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 1-Placebo: Participants aged between 12 and 17 years received eltrombopag matching placebo administered as a tablet QD for 7 weeks.
- Part 2 (Randomized Period) Cohort 1- Eltrombopag: Participants aged between 12 and 17 years received eltrombopag administered as a tablet for 7 weeks. The starting dose of eltrombopag was 37.5 mg QD. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 2-Placebo: Participants aged between 6 and 11 years received eltrombopag matching placebo administered as a tablet QD for 7 weeks.
- Part 2 (Randomized Period) Cohort 2-Eltrombopag: Participants aged between 6 and 11 years received eltrombopag administered as a tablet for 7 weeks. The starting dose of eltrombopag was based on the body weight, participants with a weight of <27 kg received 25 mg QD and participants with a weight of >=27 kg received 50 mg QD. Participants of East Asian ancestry with a body weight of <27 kg received 12.5 mg QD and participants with a weight of >=27 kg received 25 mg QD. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 3-Placebo: Participants aged between 1 to 5 years received eltrombopag matching placebo administered as a dry powder for oral suspension QD for 7 weeks.
- Part 2 (Randomized Period) Cohort 3- Eltrombopag: Participants aged between 1 to 5 years received eltrombopag administered as a dry powder for oral suspension for 7 weeks. The starting dose of eltrombopag was 1.5 mg/kg QD and the dose calculations were based on the body weight. Participants of East Asian ancestry began at 0.8 mg/kg/day. The maximum dose allowed was 2 mg/kg, unless otherwise approved by the investigator, and could not exceed 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 1: All participants aged between 12 and 17 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag starting at 37.5 mg QD up to Week 31 of the study. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 2: All participants aged between 6 and 11 years and completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag based on body weight up to Week 31 of the study. Participants with a body weight of <=27 kg received 25 mg QD and participants with a body weight of >=27 kg QD received 50 mg QD. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Open- Label Period) Cohort 3: All participants aged between 1 and 5 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag up to Week 31 of the study at 1.5 mg/kg QD. Participants of East Asian ancestry received 0.8 mg/kg/day. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Period: Part1 (24 Week Dose-Finding Period)
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3 | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Started | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 5 (Participants who completed Part 1 did not enroll in Parts 2 or 2/3) | 5 (Participants who completed Part 1 did not enroll in Parts 2 or 2/3) | 5 (Participants who completed Part 1 did not enroll in Parts 2 or 2/3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (7 Week Randomized Period)
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3 | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Started | 0 | 0 | 0 | 8 | 16 | 9 | 19 | 5 | 10 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 7 | 13 | 9 | 15 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 3 | 0 | 4 | 0 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Withdrawal by parent/ guardian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2/3(Eltrombopag Open-Label Period)
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3 | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 28 (Two participants were randomized but did not receive treatment.) | 15
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 24 (Two participants were randomized but did not receive treatment.) | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Randomized but did not receive treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Eltrombopag Dose-Finding Period: Participants (par) aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag for 24 weeks. The starting dose for Cohort 1 was 25 mg, and par of East Asian ancestry received 12.5mg QD. For Cohort 2 starting dose was based on the body weight. Par with a bodyweight of <27 kg received 12.5 mg QD, par with a body weight of >=27 kg received 25 mg QD; par of East Asian ancestry with a body weight <27 kg received 12.5 mg QD, and with a body weight of >=27 kg received 25 mg QD. For Cohort 3, the starting dose was 0.7 mg/kg QD and 0.5 mg/kg/day for par of East Asian ancestry and the dose calculations were based on the body weight. The maximum dose allowed for all Cohorts was 75mg daily. For all par, individual dose titration was allowed based upon platelet response.
- Part 2 (Randomized Period) Cohort 1-Placebo: Par aged between 12 and 17 years received eltrombopag matching placebo administered as a tablet QD for 7 weeks. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a tablet in Part 2/3. Par who received placebo in Part 2 received 24 weeks of OL treatment of eltrombopag in Part 2/3 starting at 37.5 mg QD up to Week 31 of the study. The maximum dose allowed was 75 mg daily. All par enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 1- Eltrombopag: Par aged between 12 and 17 years received eltrombopag administered as a tablet for 7 weeks. The starting dose of eltrombopag was 37.5 mg QD. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a tablet in Part 2/3. Par who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All par enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 2-Placebo: Par aged between 6 and 11 years received eltrombopag matching placebo administered as a tablet QD for 7 weeks. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a tablet in Part 2/3. Par with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Par who received placebo in Part 2 received 24 weeks of treatment of eltrombopag based on body weight up to Week 31 of the study. Par with a body weight of <=27 kg received 25 mg QD and par with a body weight of >=27 kg QD received 50 mg QD. The maximum dose allowed was 75 mg daily. All par enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 2-Eltrombopag: Par aged between 6 and 11 years received eltrombopag administered as a tablet for 7 weeks. The starting dose of eltrombopag was based on the body weight, par with a weight of <27 kg received 25 mg QD and par with a weight of >=27 kg received 50 mg QD. Par of East Asian ancestry with a body weight of <27 kg received 12.5 mg QD and par with a weight of >=27 kg received 25 mg QD. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a tablet in Part 2/3. Par with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Par who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All par enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 3-Placebo: Par aged between 1 to 5 years received eltrombopag matching placebo administered as a dry powder for oral suspension QD for 7 weeks. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Par who received placebo in Part 2 received 24 weeks of OL treatment of eltrombopag up to Week 31 of the study at 1.5 mg/kg QD. Par of East Asian ancestry received 0.8 mg/kg/day. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 3- Eltrombopag: Par aged between 1 to 5 years received eltrombopag administered as a dry powder for oral suspension for 7 weeks. The starting dose of eltrombopag was 1.5 mg/kg QD and the dose calculations were based on the body weight. Par of East Asian ancestry began at 0.8 mg/kg/day. All par completing Part 2 of the study received an OL treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Par who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All par enrolled in the study underwent individual dose titration based upon platelet response.
- Total: Total of all reporting groups
Arm/Group | Part 1 Eltrombopag Dose-Finding Period | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag | Total
Number analyzed (Participants) | 15 | 8 | 16 | 9 | 19 | 5 | 10 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.1 (4.61) | 14.6 (1.69) | 13.7 (1.58) | 8.6 (2.24) | 8.2 (1.87) | 3.6 (1.34) | 3.3 (1.34) | 9.3 (4.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 8 | 8 | 14 | 2 | 5 | 48
  Male | 7 | 5 | 8 | 1 | 5 | 3 | 5 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Asian - Japanese/East Asian Heritage | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 6
  White - White/Caucasian/European | 9 | 7 | 14 | 8 | 17 | 5 | 7 | 67
  Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White - Arabic/North African Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Mixed Race | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Platelet Count >=50 Giga Cells Per Liter (Gi/L) at Least Once, Between Day 8 and Day 43 (Weeks 1 to 6) of the Randomized Period of the Study (Part 2)
Description: Participants who achieved a platelet count >=50 Gi/L at least once between Day 8 and Day 43 (first 6 weeks of Part 2) in the absense of rescue treatment were reported. A 95% confidence interval was calculated by the exact binomial method.
Time Frame: From Day 8 up to Day 43 of Part 2
Population: Intent-to-Treat (ITT) Population: all enrolled participants during Part 2. The ITT Population was the primary population used for assessing efficacy. Only evaluable participants were considered for analysis where participants with a Baseline platelet count >10Gi/L was considered as evaluable.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 17 | 5 | 10
Percentage of Participants | 0 | 62.5 | 33.3 | 63.2 | 80.0 | 60.0

2. Secondary Outcome: Percentage of Participants Achieving Platelet Counts >=50Gi/L During Treatment With Eltrombopag in >= 60% of Assessments Between Day 15 and Day 43 (Weeks 2 Through 6) of the Randomized Treatment Period (Part 2)
Description: Sustained platelet response between the treatment groups was assessed by determining the number of participants who achieved a platelet count >=50 Gi/L during treatment with eltrombopag in >= 60% of assessments between Day 15 and Day 43 in the absence of rescue treatment were reported here.
Time Frame: Between Day 15 and Day 43 of Part 2
Population: Intent-to-Treat (ITT) Population, only those participants enrolled in Part 2 of this study were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 2 (Randomized Period) -Placebo: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag matching placebo for 7 weeks.
- Part 2 (Randomized Period) - Eltrombopag: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag for 7 weeks. The starting dose for Cohort 1 was 37.5 mg QD. For Cohort 2, starting dose was based on the body weight. Par with a body weight of <27 kg received 25 mg QD, and par with a body weight of >=27 kg received 50 mg QD. Par of East Asian ancestry with a body weight of <27 kg received 12.5 mg QD, and with a body weight of >=27 kg received 25 mg QD. For Cohort 3, the starting dose was 1.5 mg/kg QD and 0.8 mg/kg/day for par of East Asian ancestry. The maximum dose allowed was 2mg/kg and could not exceed 75 mg daily. For all par, individual dose titration was allowed based upon platelet response.
Arm/Group | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 22 | 45
Percentage of Participants | 0 | 35.6

3. Secondary Outcome: Weighted Mean Platelet Count
Description: The weighted mean platelet count is defined as the area under the platelet-time curve divided by the duration of the treatment (12 weeks). Based on the Analysis of Covariance (ANCOVA) model, the weighted mean platelet count is the sum of the Baseline count plus the age cohort plus the treatment. Baseline was defined as the platelet count taken on Day 1 or within 48 hours prior to the first dose of treatment.
Time Frame: Baseline and Day 43 of Part 2
Population: ITT Population. Only participants during Part 2 with a value at baseline and post-baseline were considered for analysis
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 21 | 43
Gi/L
  Baseline | 12.2 (8.59) | 15.5 (8.03)
  Day 43 | 30.5 (24.98) | 68 (56.78)

4. Secondary Outcome: Percentage of Participants Achieving Platelet Counts >=50Gi/L at Any Time During the 24 Weeks of Eltrombopag Dosing During Part 1.
Description: The percentage of participants achieving platelet counts >=50Gi/L at least once at any time during the 24 weeks of eltrombopag treatment were reported.
Time Frame: From Day 1 of treatment up to Week 24 of Part 1
Population: ITT Population only those participants enrolled during Part 1 were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1 (Dose-Finding Period) Cohort 1: Participants aged between 12 and 17 years received a 24-week Open-label treatment of eltrombopag administered as a tablet. The starting dose of eltrombopag was 25 milligrams (mg), once daily (QD). The participants of East Asian ancestry began at 12.5mg QD. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Percentage of Participants | 80 | 80 | 60

5. Secondary Outcome: Percentage of Participants Achieving Platelet Counts >=50 Gi/L at Any Time During the 31 Weeks of Eltrombopag Treatment During Part 2/ 3.
Description: The percentage of participants achieving platelet counts >=50Gi/L at least once at any time during the 24 weeks of eltrombopag treatment during Part 2/3 of the study were reported. Participants randmoized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: Part 2/3 up to Study Week 31
Population: ITT Population. Only evaluable participants were included for this analysis, where participants with a baseline platelet count >10 Gi/L was considered as evaluable.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 1: All participants aged between 12 and 17 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a tablet in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag starting at 37.5 mg QD up to Week 31 of the study. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 2: All participants aged between 6 and 11 years and completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag based on body weight up to Week 31 of the study. Participants with a body weight of <=27 kg received 25 mg QD and participants with a body weight of >=27 kg QD received 50 mg QD. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 3: All participants aged between 1 and 5 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag up to Week 31 of the study at 1.5 mg/kg QD. Participants of East Asian ancestry received 0.8 mg/kg/day. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Percentage of Participants | 75.0 | 82.1 | 86.7

6. Secondary Outcome: Population Pharmacokinetic (PK) Assessment for Eltrombopag for AUC(0-t) During Part 1, 2, and 2/3.
Description: The area under the concentration-time curve over the dosing interval (AUC0-t) data was collected to estimate primary model-based PK parameters. PK samples were collected within 3 hours prior to dosing and 2, 4, 6, 8 and 24 hours after dosing. Doses were normalized to 50mg for comparison. PK samples were collected at each on-treatment visit during Part 1, Part 2, and Part 2/3. The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. AUC(0-t) is defined as the area under the concentration-time curve over the dosing interval. From the final model, a single value of AUC(0-t) was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: From Day 1 of treatment up to Study Week 31
Population: Pharmacokinetic (PK) population. All subjects who had received at least one dose of the investigational product and provided a PK sample were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram*hour per milliliter (ug*h/mL)
Groups:
- Eltrombopag Cohort 1- 12-17 Years: Participants (par) aged between 12 and 17 years received eltrombopag administered as a tablet for a total of 24 weeks. Par in Part 1 received an Open-Label (OL) treatment (trt) starting at 25 milligrams (mg) once daily (QD) for 24 weeks. Par of East Asian ancestry began at 12.5mg QD. Par randomized to eltrombopag in Part 2 received eltrombopag for 7 weeks starting at 37.5mg QD. All par completing Part 2 received an OL trt of eltrombopag in Part 2/3. Par who received 7 weeks of eltrombopag in Part 2 received an additional 17 weeks of trt to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. Par who received placebo Part 2, received 24 weeks of trt of eltrombopag in Part 2/3 starting at 37.5 mg QD up to Week 31 of the study. The maximum dose allowed was 75mg daily. All par underwent individual dose titration based upon platelet response.
- Eltrombopag Cohort 2 - 6-11 Years: Par aged between 6 and 11 years received eltrombopag administered as a tablet or dry powder for oral suspension for a total of 24 weeks. Par in Part 1 received an OL trt based on body weight for 24 weeks. Par weighing <27 kilograms (kg) started at 12.5mg QD and par weighing >=27kg started at 25mg QD. Par randomized to eltrombopag in Part 2 received trt based on body weight for 7 weeks. Par weighing <27kg started at 25mg QD and par weighing >=27kg started at 50mg QD. Par of East Asian ancestry weighing <27kg began at 12.5mg QD and those >=27kg began at 25mg QD. Par who received 7 weeks of eltrombopag in Part 2 continued the same dose in Part 2/3 for an additional 17 weeks of trt to complete a total of 24 weeks. Par who received placebo in Part 2, received 24 weeks of trt of eltrombopag in Part 2/3 using the same dosing guidelines as Part 2 up to Week 31 of the study. The maximum dose allowed was 75mg daily. All par underwent individual dose titration based upon platelet response.
- Eltrombopag Cohort 3 - 1-5 Years: Par aged between 1 and 5 years received eltrombopag administered as a dry powder for oral suspension for a total of 24 weeks. Par in Part 1 received an OL trt based on body weight for 24 weeks. Par starting dose was 0.7mg/kg QD, par of East Asian ancestry began at 0.5mg/kg/day. Par randomized to eltrombopag in Part 2 received trt based on body weight for 7 weeks. Par starting dose was 1.5mg/kg QD, par of East Asian ancestry weighing began at 0.8 mg/kg/day. Par who received 7 weeks of eltrombopag in Part 2 continued the same dose in Part 2/3 for an additional 17 weeks of trt to complete a total of 24 weeks. Par who received placebo in Part 2, received 24 weeks of trt of eltrombopag in Part 2/3 using the same dosing guidelines as Part 2 up to Week 31 of the study. The maximum dose allowed was 75mg daily. All par underwent individual dose titration based upon platelet response.
Arm/Group | Eltrombopag Cohort 1- 12-17 Years | Eltrombopag Cohort 2 - 6-11 Years | Eltrombopag Cohort 3 - 1-5 Years
Number analyzed (Participants) | 29 | 30 | 19
Microgram*hour per milliliter (ug*h/mL) | 101 [87.1 to 117] | 132 [114 to 152] | 142 [117 to 173]

7. Secondary Outcome: Population Pharmacokinetic (PK) Assessments for Eltrombopag for Cmax and Ct During Part 1, 2, and 2/3.
Description: The maximum observed concentration (Cmax) and the concentration at the end of the dosing interval (Ct) data were collected to estimate primary model-based PK parameters. PK samples were collected within 3 hours prior to dosing and 2, 4, 6, 8 and 24 hours after dosing. Doses were normalized to 50mg for comparison. PK samples were collected at each on-treatment visit during Part 1, Part 2, and Part 2/3. The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. From the final model, a single value of Cmax and Ct were estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: From Day 1 of treatment up to Study Week 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (ug/mL)
Arm/Group | Eltrombopag Cohort 1- 12-17 Years | Eltrombopag Cohort 2 - 6-11 Years | Eltrombopag Cohort 3 - 1-5 Years
Number analyzed (Participants) | 29 | 30 | 19
micrograms per milliliter (ug/mL)
  Cmax | 6.65 [5.87 to 7.53] | 9.19 [8.18 to 10.3] | 10.7 [9.24 to 12.5]
  Ct | 2.42 [1.97 to 2.98] | 2.95 [2.41 to 3.60] | 2.91 [2.14 to 3.96]

8. Secondary Outcome: Population Pharmacokinetic (PK) Assessments for Eltrombopag for Tmax During Part 1, 2, and 2/3
Description: The time to maximum concentration (tmax) was collected to estimate primary model-based PK parameters. PK samples were collected within 3 hours prior to dosing and 2, 4, 6, 8 and 24 hours after dosing. PK samples were collected at each on-treatment visit during Part 1, Part 2, and Part 2/3. The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. From the final model, a single value of tmax was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: From Day 1 of treatment up to Study Week 31
Population: as for outcome 6
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Eltrombopag Cohort 1- 12-17 Years | Eltrombopag Cohort 2 - 6-11 Years | Eltrombopag Cohort 3 - 1-5 Years
Number analyzed (Participants) | 29 | 30 | 19
hour (hr) | 4.0 [2.0 to 6.0] | 4.0 [2.0 to 6.0] | 2.0 [2.0 to 4.0]

9. Secondary Outcome: Population Pharmacokinetic (PK) Assessments for Eltrombopag for CL/F During Part 1, 2, and 2/3
Description: The apparent plasma clearance following oral dosing of eltrombopag (CL/F) was collected to estimate primary model-based PK parameters. PK samples were collected within 3 hours prior to dosing and 2, 4, 6, 8 and 24 hours after dosing. PK samples were collected at each on-treatment visit during Part 1, Part 2, and Part 2/3. The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. From the final model, a single value of CL/F was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: From Day 1 of treatment up to Study Week 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: liter per hour (L/hr)
Arm/Group | Eltrombopag Cohort 1- 12-17 Years | Eltrombopag Cohort 2 - 6-11 Years | Eltrombopag Cohort 3 - 1-5 Years
Number analyzed (Participants) | 29 | 30 | 19
liter per hour (L/hr) | 0.50 [0.43 to 0.57] | 0.38 [0.33 to 0.44] | 0.25 [0.20 to 0.30]

10. Secondary Outcome: Maximum Duration for Which a Participant Continuously Maintained a Platelet Count of >=50 Gi/L During the 7 Weeks of Eltrombopag Treatment in Part 2
Description: The maximum duration for which a participant continuously maintained a platelet count >=50 Gi/L in the absence of rescue treatment was calculated and summarized during the 24 weeks of eltrombopag treatment in Part 2. Participants with non-weekly assessments were assumed to have maintained a positive response for each week between two assessments that had positive responses. If a particpant achieved a positive response at an assessment and then achieved a negative response at the next assessment, then it was assumed that the participant had achieved a positive response for one day. Excludes periods from initiation of rescue medication until platelet count falls to below 50Gi/L, irrespective of platelet count
Time Frame: From Baseline through Week 7 of Part 2
Population: ITT Population, only those participants enrolled in Part 2 were analyzed. The number of participants used to compute the summary statistics reflect the ITT poplation through out the analyses during Part 2.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 19 | 5 | 10
Weeks | 0.0 [0 to 0] | 1.0 [0 to 5] | 0.0 [0 to 2] | 2.0 [0 to 6] | 1.0 [0 to 2] | 1.0 [0 to 6]

11. Secondary Outcome: Maximum Duration for Which a Participant Continuously Maintained a Platelet Count of >=50 Gi/L During the 24 Weeks of Eltrombopag Treatment in Part 2/ 3
Description: The maximum duration for which a participant continuously maintained a platelet count >=50 Gi/L in the absence of rescue treatment was calculated and summarized during the 24 weeks of eltrombopag treatment in Part 2/3. Participants with non-weekly assessments were assumed to have maintained a positive response for each week between two assessments that had positive responses. If a particpant achieved a positive response at an assessment and then achieved a negative response at the next assessment, then it was assumed that the participant had achieved a positive response for one day. Participants randmoized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: From Baseline up to Study Week 31
Population: ITT Population only those participants enrolled in Part 2/3 were analyzed. The number of participants used to compute the summary statistics reflect the ITT poplation through out the analyses during Part 2/3.
Measure: Median (Full Range); unit: Weeks
Groups:
- Part 2/3 (Eltrombopag Open-Label Period) Cohort 3: All participants aged between 1 and 5 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag up to Week 31 of the study at 1.5 mg/kg QD. Participants of East Asian ancestry received 0.8 mg/kg/day. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 3
Number analyzed (Participants) | 24 | 28 | 15
Weeks | 2.0 [0 to 23] | 8.0 [0 to 24] | 4.0 [0 to 24]

12. Secondary Outcome: Percentage of Participants Who Reduced or Discontinued Baseline Concomitant Idiopathic Thrombocytopenic Purpura (ITP) Medications During the 24 Weeks of Eltrombopag Treatment During Part 1.
Description: The participants who discontinued (dis) or had a sustained reduction (red) of a Baseline (BL) ITP medication for at least one day during the period of Day 1 of Part 1 to the last dose of study medication +1 day are reported. The denominator is the number of subjects taking an ITP medication at baseline. For participants in Part 1, Baseline is defined as Day 1 of Part 1. A sustained reduction is defined as reduction for 4 weeks or more. An attempted red or dis is a decrease in the dose or frequency from the BL dose or frequency of an ITP medication for at least one day during the period Part 1 Day 1 to the last dose of study medication + 1 day.
Time Frame: From Baseline up to Week 24+ 1 day of Part 1
Population: ITT Population, only those participants enrolled during Part 1 were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Percentage of Participants
  Taking an ITP medication at BL | 0 | 20.0 | 0
  Attempted red or dis | 0 | 100.0 | 0
  Permanent red or dis of all BL ITP mediation | 0 | 100.0 | 0
  Permanent red or dis at least 1 BL ITP medcation | 0 | 100.0 | 0

13. Secondary Outcome: Percentage of Participants Who Reduced or Discontinued Baseline Concomitant ITP Medications During the 24 Weeks of Eltrombopag Treatment During Part 2/ 3
Description: Participants who discontinued (dis) or had a sustained reduction (red) of a Baseline (BL) ITP medication for at least one day during the period of Day 1 of Part 2/3 to the last dose of study medication +1 day are reported. The denominator is the number of subjects taking an ITP medication at baseline. For participants randomized to placebo in Part 2, BL is defined as Week 7 of Part 2. For participants randomized to eltrombopag in Part 2, BL is defined as Day 1 of Part 2. A sustained reduction is defined as reduction for 4 weeks or more. An attempted reduction or discontinuation is a decrease in the dose or frequency from the BL dose or frequency of an ITP medication for at least one day during the period Part 2/3 Day 1 to the last dose of study medication + 1 day.
Time Frame: From Baseline to the end of treatment up to Week 31 + 1 day of Part 2/3
Population: ITT Population, only those participants enrolled during Part 2/3 were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 3
Number analyzed (Participants) | 24 | 28 | 15
Percentage of Participants
  Taking an ITP medication at BL | 25.0 | 17.9 | 13.3
  Attempted red or dis | 66.7 | 20.0 | 100.0
  Permanent (perm) dis of all BL ITP medication(med) | 16.7 | 20.0 | 50.0
  Perm dis at least 1 BL ITP med | 33.3 | 20.0 | 50.0
  Perm dis all BL ITP med taken prior to Part 2/3 | 0 | 40.0 | 0

14. Secondary Outcome: Number of Participants Who Required a Protocol-defined Rescue Treatment During Part 2/3
Description: Rescue treatment was defined as either a new immune (idiopathic) thrombocytopenic purpura (ITP) medication, an increase in the dose of a concomitant ITP medication from Baseline, a platelet transfusion, or a splenectomy. For particpants randomized to placebo in Part 2, Baseline is defined as Week 7 of Part 2. For participants randomized to eltrombopag in Part 2, Baseline is defined as Day 1 of Part 2. Participants randmoized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: From Baseline to the end of treatment up to Week 31 + 1 day of Part2/3
Population: ITT Population, only those participants enrolled during Part 2/3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 3
Number analyzed (Participants) | 24 | 28 | 15
Participants
  New ITP Medication | 8 | 4 | 4
  Increase concomitant ITP medication from Baseline | 1 | 0 | 0
  Platelet transfusion | 0 | 0 | 0
  Splenectomy | 0 | 0 | 0

15. Secondary Outcome: Kids' ITP Tool (KIT) Questionnaire Total Score at Baseline, Week 6, Week 12, and Week 24 as Assessed Using the KIT Questionnaire During the Dose Finding Period, Part 1
Description: The KIT questionnaire measures the impact on the quality of life determined by the participant and the guardian by self reported outcomes at Baseline or the Screening Visit, after 6 weeks of treatment, after 12 weeks of treatment and at the end of treatment or withdrawal from the study. The KIT total score is calculated from the scores of each of the individual questions from Q1 - Q26 (excluding any answer that is 'Not applicable'). The code list used for the individual question scores is: 1 = never, 2 = seldom, 3 = sometimes, 4 = often, 5 = always and 9 = not applicable. The range of values the total score can take is 0 (worst) to 100 (best). For subjects under the age of six, the family questionnaire (parental proxy) has been used.
Time Frame: Baseline, Week 6, Week 12, and Week 24 of Part 1
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Score on scale
  Baseline, n=5, 5, 5 | 73.18 (15.743) | 53.95 (16.534) | 74.80 (17.199)
  Week 6, n=4, 5, 5 | 82.84 (9.131) | 61.57 (13.664) | 71.54 (14.798)
  Week 12, n=4, 4, 4 | 84.14 (11.712) | 66.43 (12.349) | 65.58 (17.887)
  Week 24, n= 3, 4, 3 | 76.38 (20.228) | 82.50 (15.995) | 78.87 (12.056)

16. Secondary Outcome: Kids' ITP Tool (KIT) Questionnaire Total Score at Baseline and Week 6as Assessed Using the KIT Questionnaire During the Randomized Period, Part 2
Description: The KIT questionnaire measures the impact on the quality of life determined by the participant and the guardian by self reported outcomes at Baseline or the Screening Visit, after 6 weeks of treatment or withdrawal from the study. The KIT total score is calculated from the scores of each of the individual questions from Q1 - Q26 (excluding any answer that is 'Not applicable'). The code list used for the individual question scores is: 1 = never, 2 = seldom, 3 = sometimes, 4 = often, 5 = always and 9 = not applicable. The range of values the total score can take is 0 (worst) to 100 (best). For subjects under the age of six, the family questionnaire (parental proxy) has been used.
Time Frame: Baseline and Week 6 of Part 2
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 19 | 5 | 10
Score on scale
  Baseline, n=6, 11, 9, 10, 2, 8 | 83.94 (8.674) | 76.84 (15.049) | 71.05 (19.581) | 66.36 (17.321) | 82.61 (7.686) | 78.23 (9.575)
  Week 6, n= 8,11,7,13, 5, 9 | 79.46 (10.971) | 79.46 (13.899) | 74.65 (20.968) | 80.16 (13.776) | 88.01 (3.333) | 80.85 (15.082)

17. Secondary Outcome: Kids' ITP Tools (KIT) Questionnaire Total Score at Baseline, Week, 6, Week 12, and End of Treatment Visit as Assessed Using the KIT Questionnaire During the Eltrombopag Open-Label Period, Part 2/3
Description: The KIT questionnaire measures the impact on the quality of life determined by the participant and the guardian by self reported outcomes at Baseline or the Screening Visit, after 6 weeks of treatment, after 12 weeks of treatment and at the end of treatment or withdrawal from the study. The KIT total score is calculated from the scores of each of the individual questions from Q1 - Q26 (excluding any answer that is 'Not applicable'). The code list used for the individual question scores is: 1=never, 2=seldom, 3=sometimes, 4=often, 5=always and 9=not applicable. The range of values the total score can take is 0 (worst) to 100 (best). For subjects under the age of six, the family questionnaire (parental proxy) has been used.
Time Frame: From Baseline to end of treatment up to Study Week 31
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Part 2/3 (Eltrombopag Period) Cohort 1: All participants aged between 12 and 17 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag starting at 37.5 mg QD up to Week 31 of the study. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Period) Cohort 2: All participants aged between 6 and 11 years and completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag based on body weight up to Week 31 of the study. Participants with a body weight of <=27 kg received 25 mg QD and participants with a body weight of >=27 kg QD received 50 mg QD. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Period) Cohort 3: All participants aged between 1 and 5 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Participants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag up to Week 31 of the study at 1.5 mg/kg QD. Participants of East Asian ancestry received 0.8 mg/kg/day. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 2/3 (Eltrombopag Period) Cohort 1 | Part 2/3 (Eltrombopag Period) Cohort 2 | Part 2/3 (Eltrombopag Period) Cohort 3
Number analyzed (Participants) | 24 | 28 | 15
Score on scale
  Baseline, n=17, 18, 10 | 79.34 (13.315) | 70.59 (16.237) | 79.10 (9.016)
  Week 6, n=11, 13, 9 | 79.46 (13.899) | 80.16 (13.776) | 80.85 (15.082)
  Week 12, n=9, 7, 2 | 84.25 (7.531) | 76.48 (19.948) | 88.10 (11.166)
  Week 24, n=17, 11, 8 | 82.16 (16.926) | 83.93 (13.327) | 77.93 (22.971)

18. Secondary Outcome: Number of Participants With Any Bleeding, no Clinically Significant Bleeding and Significant Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale During Part 2
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: Grade 0 = no bleeding, Grade 1 = petechiae, Grade 2 = mild blood loss, Grade 3 = gross bleeding and Grade 4 = debilitating blood loss. The WHO grades were dichotomized into the following categories: no bleeding=Grade 0; any bleeding=Grades 1 to 4; no clinically significant bleeding=Grades 0 to 1; clinically significant bleeding=Grades 2 to 4. For participants randomized to Placebo in Part 2, Baseline defined as Week 7 of Part 2. For participants randomized to Eltrombopag in Part 2, Baseline defined as Day 1 of Part 2.
Time Frame: From Baseline through Week 7 of Part 2
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 19 | 5 | 10
Participants
  Baseline, Grades 1-4, n=8, 16, 9, 19, 5, 10 | 6 | 16 | 7 | 11 | 5 | 8
  Baseline, Grades 0-1, n=8, 16, 9, 19, 5, 10 | 6 | 13 | 6 | 17 | 4 | 6
  Baseline, Grades 2-4, n=8, 16, 9, 19, 5, 10 | 2 | 3 | 3 | 2 | 1 | 4
  Week 1, Grades 1-4, n=8, 16, 9, 17, 5, 10 | 7 | 9 | 6 | 7 | 3 | 7
  Week 1, Grades 0-1, n=8, 16, 9, 17, 5, 10 | 3 | 14 | 6 | 17 | 5 | 5
  Week 1, Grades 2-4, n=8, 16, 9, 17, 5, 10 | 5 | 2 | 3 | 0 | 0 | 5
  Week 2, Grades 1-4, n=8, 16, 9, 17, 5, 10 | 7 | 11 | 6 | 6 | 2 | 5
  Week 2, Grades 0-1, n=8, 16, 9, 17, 5, 10 | 5 | 13 | 7 | 16 | 3 | 7
  Week 2, Grades 2-4, n=8, 16, 9, 17, 5, 10 | 3 | 3 | 2 | 1 | 2 | 3
  Week 3, Grades 1-4, n=8, 16, 9, 16, 5, 9 | 6 | 10 | 7 | 6 | 2 | 5
  Week 3, Grades 0-1, n=8, 16, 9, 16, 5, 9 | 5 | 14 | 7 | 14 | 3 | 7
  Week 3, Grades 2-4, n=8, 16, 9, 16, 5, 9 | 3 | 2 | 2 | 2 | 2 | 2
  Week 4, Grades 1-4, n=8, 16, 9, 17, 5, 9 | 6 | 7 | 7 | 7 | 2 | 6
  Week 4, Grades 0-1, n=8, 16, 9, 17, 5, 9 | 6 | 16 | 8 | 17 | 3 | 7
  Week 4, Grades 2-4, n=8, 16, 9, 17, 5, 9 | 2 | 0 | 1 | 0 | 2 | 2
  Week 5, Grades 1-4, n=8, 16, 9, 16, 5, 9 | 6 | 8 | 7 | 3 | 4 | 5
  Week 5, Grades 0-1, n=8, 16, 9, 16, 5, 9 | 4 | 14 | 8 | 16 | 4 | 8
  Week 5, Grades 2-4, n=8, 16, 9, 16, 5, 9 | 4 | 2 | 1 | 0 | 1 | 1
  Week 6, Grades 1-4, n=8, 16, 9, 17, 5, 9 | 5 | 2 | 7 | 4 | 4 | 4
  Week 6, Grades 0-1, n=8, 16, 9, 17, 5, 9 | 7 | 16 | 7 | 16 | 4 | 9
  Week 6, Grades 2-4, n=8, 16, 9, 17, 5, 9 | 1 | 0 | 2 | 1 | 1 | 0
  Week 7, Grades 1-4, n=8, 16, 9, 17, 5, 9 | 7 | 5 | 7 | 5 | 4 | 4
  Week 7, Grades 0-1, n=8, 16, 9, 17, 5, 9 | 4 | 15 | 8 | 16 | 3 | 7
  Week 7, Grades 2-4, n=8, 16, 9, 17, 5, 9 | 4 | 1 | 1 | 1 | 2 | 2

19. Secondary Outcome: Number of Participants With Any Bleeding, no Clinically Significant Bleeding and Significant Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale During Part 2/3
Description: as for outcome 18
Time Frame: From Baseline of Part 2/3 through Follow-up
Population: as for outcome 15
Measure: Number; unit: Participants
Groups:
- Part 2/ 3 (Eltrombopag Period) Cohort 1: All participants aged between 12 and 17 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a tablet in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag starting at 37.5 mg QD up to Week 31 of the study. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Period) Cohort 2: All participants aged between 6 and 11 years and completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet in Part 2/3. Participants with difficulty swallowing a tablet in Part 2 were administered eltrombopag as a dry powder for oral suspension in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag based on body weight up to Week 31 of the study. Participants with a body weight of <=27 kg received 25 mg QD and participants with a body weight of >=27 kg QD received 50 mg QD. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2/3 (Eltrombopag Period) Cohort 3: All participants aged between 1 and 5 years and completing Part 2 of the study received an Open-Label treatment of eltrombopag administered as a dry powder for oral suspension in Part 2/3. Particpiants who received placebo in Part 2 received 24 weeks of treatment of eltrombopag up to Week 31 of the studyat 1.5 mg/kg QD. Participants of East Asian ancestry received 0.8 mg/kg/day. Participants who received 7 weeks of eltrombopag treatment in Part 2 received an additional 17 weeks of treatment to complete a total of 24 weeks continuing at the same dosage at the end of Part 2. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 2/ 3 (Eltrombopag Period) Cohort 1 | Part 2/3 (Eltrombopag Period) Cohort 2 | Part 2/3 (Eltrombopag Period) Cohort 3
Number analyzed (Participants) | 24 | 28 | 15
Participants
  Baseline, Grades 1-4, n=24, 28, 15 | 23 | 18 | 12
  Baseline, Grades 0-1, n=24, 28, 15 | 17 | 25 | 9
  Baseline, Grades 2-4, n=24, 28, 15 | 7 | 3 | 6
  Week 1, Grades 1-4, n=24, 26, 15 | 14 | 13 | 9
  Week 1, Grades 0-1, n=24, 26, 15 | 20 | 24 | 9
  Week 1, Grades 2-4, n=24, 26, 15 | 4 | 2 | 6
  Week 2, Grades 1-4, n=24, 26, 14 | 15 | 12 | 8
  Week 2, Grades 0-1, n=24, 26, 14 | 21 | 23 | 10
  Week 2, Grades 2-4, n=24, 26, 14 | 3 | 3 | 4
  Week 3, Grades 1-4, n=24, 25, 14 | 13 | 9 | 6
  Week 3, Grades 0-1, n=24, 25, 14 | 21 | 23 | 12
  Week 3, Grades 2-4, n=24, 25, 14 | 3 | 2 | 2
  Week 4, Grades 1-4, n=24, 26, 13 | 10 | 11 | 8
  Week 4, Grades 0-1, n=24, 26, 13 | 24 | 26 | 10
  Week 4, Grades 2-4, n=24, 26, 13 | 0 | 0 | 3
  Week 5, Grades 1-4, n=24, 24, 13 | 11 | 4 | 9
  Week 5, Grades 0-1, n=24, 24, 13 | 21 | 24 | 12
  Week 5, Grades 2-4, n=24, 24, 13 | 3 | 0 | 1
  Week 6, Grades 1-4, n=23, 24, 12 | 6 | 6 | 4
  Week 6, Grades 0-1, n=23, 24, 12 | 23 | 22 | 12
  Week 6, Grades 2-4, n=23, 24, 12 | 0 | 2 | 0
  Week 7, Grades 1-4, n=22, 25, 14 | 8 | 7 | 4
  Week 7, Grades 0-1, n=22, 25, 14 | 20 | 24 | 12
  Week 7, Grades 2-4, n=22, 25, 14 | 2 | 1 | 2
  Week 8, Grades 1-4, n=19, 21, 11 | 10 | 6 | 5
  Week 8, Grades 0-1, n=19, 21, 11 | 19 | 19 | 9
  Week 8, Grades 2-4, n=19, 21, 11 | 0 | 2 | 2
  Week 9, Grades 1-4, n=17, 16, 12 | 8 | 5 | 6
  Week 9, Grades 0-1, n=17, 16, 12 | 13 | 16 | 10
  Week 9, Grades 2-4, n=17, 16, 12 | 4 | 0 | 2
  Week 10, Grades 1-4, n=16, 14, 11 | 5 | 5 | 7
  Week 10, Grades 0-1, n=16, 14, 11 | 16 | 12 | 11
  Week 10, Grades 2-4, n=16, 14, 11 | 0 | 2 | 0
  Week 11, Grades 1-4, n=16, 15, 12 | 15 | 5 | 7
  Week 11, Grades 0-1, n=16, 15, 12 | 16 | 13 | 10
  Week 11, Grades 2-4, n=16, 15, 12 | 0 | 2 | 2
  Week 12, Grades 1-4, n=19, 16, 9 | 6 | 7 | 4
  Week 12, Grades 0-1, n=19, 16, 9 | 18 | 14 | 7
  Week 12, Grades 2-4, n=19, 16, 9 | 1 | 2 | 2
  Week 13, Grades 1-4, n=12, 14, 10 | 6 | 5 | 6
  Week 13, Grades 0-1, n=12, 14, 10 | 12 | 13 | 10
  Week 13, Grades 2-4, n=12, 14, 10 | 0 | 1 | 0
  Week 14, Grades 1-4, n=15, 11, 17 | 3 | 2 | 3
  Week 14, Grades 0-1, n=15, 11, 17 | 15 | 11 | 5
  Week 14, Grades 2-4, n=15, 11, 17 | 0 | 0 | 2
  Week 15, Grades 1-4, n=12, 14, 6 | 6 | 3 | 3
  Week 15, Grades 0-1, n=12, 14, 6 | 10 | 14 | 5
  Week 15, Grades 2-4, n=12, 14, 6 | 2 | 0 | 1
  Week 16, Grades 1-4, n=17, 15, 9 | 7 | 8 | 4
  Week 16, Grades 0-1, n=17, 15, 9 | 17 | 14 | 9
  Week 16, Grades 2-4, n=17, 15, 9 | 0 | 1 | 0
  Week 17, Grades 1-4, n=13, 11, 5 | 5 | 3 | 4
  Week 17, Grades 0-1, n=13, 11, 5 | 13 | 11 | 5
  Week 17, Grades 2-4, n=13, 11, 5 | 0 | 0 | 0
  Week 18, Grades 1-4, n=16, 12 ,4 | 3 | 2 | 3
  Week 18, Grades 0-1, n=16, 12 ,4 | 16 | 11 | 4
  Week 18, Grades 2-4, n=16, 12 ,4 | 0 | 1 | 0
  Week 19, Grades 1-4, n=14, 15, 7 | 3 | 4 | 1
  Week 19, Grades 0-1, n=14, 15, 7 | 14 | 14 | 7
  Week 19, Grades 2-4, n=14, 15, 7 | 0 | 1 | 0
  Week 20, Grades 1-4, n=13, 13, 8 | 2 | 3 | 2
  Week 20, Grades 0-1, n=13, 13, 8 | 13 | 13 | 6
  Week 20, Grades 2-4, n=13, 13, 8 | 0 | 0 | 2
  Week 21, Grades 1-4, n=4, 10, 3 | 1 | 0 | 0
  Week 21, Grades 0-1, n=4, 10, 3 | 4 | 10 | 3
  Week 21, Grades 2-4, n=4, 10, 3 | 0 | 0 | 0
  Week 22, Grades 1-4, n=12,7, 5 | 2 | 2 | 2
  Week 22 Grades 0-1, n=12,7, 5 | 12 | 6 | 5
  Week 22 Grades 2-4, n=12,7, 5 | 0 | 1 | 0
  Week 23, Grades 1-4, n=8, 7,6 | 1 | 1 | 2
  Week 23, Grades 0-1, n=8, 7,6 | 8 | 7 | 6
  Week 23, Grades 2-4, n=8, 7,6 | 0 | 0 | 0
  Week 24, Grades 1-4, n=23, 24, 13 | 5 | 5 | 4
  Week 24, Grades 0-1, n=23, 14, 13 | 21 | 24 | 12
  Week 24, Grades 2-4, n=23, 14, 13 | 2 | 0 | 1
  Follow Up Week 1, Grades 1-4, n=8, 5, 3 | 5 | 1 | 3
  Follow Up Week 1, Grades 0-1, n=8, 5, 3 | 8 | 4 | 2
  Follow Up Week 1, Grades 2-4, n=8, 5, 3 | 0 | 1 | 1
  Follow Up Week 2, Grades 1-4, n=7, 7, 7 | 2 | 6 | 2
  Follow Up Week 2, Grades 0-1, n=7, 7, 7 | 7 | 6 | 6
  Follow Up Week 2, Grades 2-4, n=7, 7, 7 | 0 | 1 | 1
  Follow Up Week 3, Grades 1-4, n=5, 5, 5 | 1 | 2 | 4
  Follow Up Week 3, Grades 0-1, n=5, 5, 5 | 5 | 5 | 4
  Follow Up Week 3, Grades 2-4, n=5, 5, 5 | 0 | 0 | 1
  Follow Up Week 4, Grades 1-4, n=9, 14, 8 | 5 | 4 | 3
  Follow Up Week 4, Grades 0-1, n=9, 14, 8 | 8 | 13 | 7
  Follow Up Week 4, Grades 2-4, n=9, 14, 8 | 1 | 1 | 1
  Any Follow Up Visit, Grades 1, n=15, 18, 10 | 7 | 10 | 5
  Any Follow Up Visit, Grades 0-1, n=15, 18, 10 | 15 | 18 | 9
  Any Follow Up Visit, Grades 2-4, n=15, 18, 10 | 1 | 3 | 3

20. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Parameter Falling Outside of the Reference Range Any Time Post-Baseline During Part 1, Part 2, and Part 2/3
Description: Clinical chemistry parameters included: aspartate amino transferase (AST, reference range [RR]: 0-38 International Units per Liter [IU/L]), alkaline phosphatase (ALP: RR: 50 - 375 IU/L), total bilirubin (RR: 3.42 - 22.23 micromoles [umol]/L), albumin grams [g/L], alanine amino transferase (ALT, RR: 5-30 IU/L), prothrombin international normalized ratio (PT INR, RR-0.9 - 1.2), activated partial thromboplastin time (APTT, RR: 24.2 - 32.9 seconds), glucose (RR: 4.107- 6.55018 millimoles [mmol]/L), potassium (3 - 5 mmol/L), and sodium (135 - 143 mmol/L). Baseline values were obtained at Day 1. The number of participants with the indicated clinical chemistry data outside of the reference range (with high and low) any time post-Baseline are presented. Anytime post-Baseline assesments included any scheduled and unscheduled post-Baseline assessment
Time Frame: Post-Baseline from Week 1 through Follow-up up to Study Week 35
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Groups:
- Part 1 (Dose-Finding Period): Participants (par) aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag for 24 weeks. The starting dose for Cohort 1 was 25 mg, and par of East Asian ancestry received 12.5mg QD. For cohort 2 starting dose was based on the body weight. Par with a body weight of <27 kg received 12.5 mg QD, par with a body weight of >=27 kg received 25 mg QD; par of east Asian ancestry with a body weight <27 kg received 12.5 mg QD, and with a body weight of >=27 kg received 25 mg QD. For Cohort 3, the starting dose was 0.7 mg/kg QD and 0.5 mg/kg/day for par of East Asian ancestry and the dose calculations were based on the body weight. The maximum dose allowed for all Cohorts was 75mg daily. For all par, individual dose titration was allowed based upon platelet response.
- Part 2/3 (Eltrombopag Open-Label Period): Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3: 1 to 5 years), completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet or dry powder for oral suspension in Part 2/3. Par who received eltrombopag during the Randomized Period continued on the same dose, unless adjustments were warranted according to the dosing guidelines, for 17 additional weeks (for a total of 24 weeks of treatment). Par who received placebo during the Randomized Period followed the starting doses for each age Cohort specified for Part 2, and received a total of 24 weeks of eltrombopag treatment.
Arm/Group | Part 1 (Dose-Finding Period) | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag | Part 2/3 (Eltrombopag Open-Label Period)
Number analyzed (Participants) | 15 | 21 | 44 | 65
Participants
  AST high, n=15, 21, 44, 65 | 5 | 4 | 7 | 17
  AST low, n=15, 21, 44, 65 | 1 | 1 | 3 | 7
  ALT, high, n= 15, 21, 44, 65 | 2 | 3 | 3 | 14
  ALT, low, n= 15, 21, 44, 65 | 2 | 3 | 4 | 11
  Total Bilirubin, high, n=15, 21, 44, 65 | 5 | 2 | 2 | 9
  Total Bilirubin, low, n=15, 21, 44, 65 | 6 | 0 | 16 | 31
  Direct Bilirubin, high, n=10, 16, 34, 55 | 0 | 1 | 1 | 3
  Direct Bilirubin, low, n=10, 16, 34, 55 | 1 | 0 | 6 | 8
  Albumin, high, n=15, 21, 24, 65 | 3 | 3 | 2 | 9
  Albumin, low, n=15, 21, 24, 65 | 1 | 3 | 5 | 11
  ALP, high, n=15, 21, 24, 65 | 4 | 1 | 6 | 13
  ALP, low, n=15, 21, 24, 65 | 2 | 2 | 4 | 11
  PT INR, high, n=15, 20, 42, 64 | 2 | 1 | 4 | 12
  PT INR, low, n=15, 20, 42, 64 | 0 | 0 | 0 | 1
  PT, high, n=13, 20, 36, 61 | 5 | 5 | 8 | 24
  PT, low, n=13, 20, 36, 61 | 0 | 1 | 0 | 3
  PTT, high, n=15, 21, 41, 63 | 4 | 2 | 1 | 11
  PTT, low, n=15, 21, 41, 63 | 0 | 1 | 1 | 9
  Glucose, high, n=15, 21, 44, 65 | 5 | 5 | 7 | 27
  Glucose, low, n=15, 21, 44, 65 | 7 | 6 | 16 | 29
  Potassium, high, n=15, 21, 44, 65 | 7 | 0 | 3 | 9
  Potassium, low, n=15, 21, 44, 65, | 3 | 4 | 8 | 14
  Sodium, high, n=15, 21, 44, 65 | 2 | 1 | 2 | 6
  Sodium, low, n=15, 21, 44, 65 | 2 | 1 | 4 | 9

21. Secondary Outcome: Number of Participants With the Indicated Hematology Parameters Falling Outside of the Reference Range at Any Time Post-Baseline During Part 1, Part 2, and Part 2/3
Description: Hematology parameters included: erythrocytes (RR: 4.2 - 6.1 teragrams per liter [TI/L]), hemoglobin (RR: 125 - 165 g/L), hematocrit (RR: 0.36 - 0.46), platelets (RR: 170 - 430 gigagrams per liter [GI/L]), mean platelet volume (MPV, RR: 4 - 14 femotoliter [fL]), leukocytes (RR: 3.4 - 11.2 GI/L), total neutrophils (RR: 2.1 - 4.9 GI/L), lymphocytes (RR: 1.4 - 2.9 GI/L), monocytes (RR: 0.2 - 0.9 GI/L), eosinophils (RR: 0.2 - 0.7 GI/L), and basophils (RR: 0.02 - 0.12 GI/L). Baseline values were obtained at Day 1. The number of participants with the indicated hematology parameters data outside of the reference range (with high and low) any time post-baseline are presented. Anytime post-Baseline assesments included any scheduled and unscheduled post-Baseline assessment
Time Frame: Post-Baseline from Week 1 through Follow-up up to Study Week 35
Population: as for outcome 20
Measure: Number; unit: Participants
Groups:
- Part 1 (Dose-Finding Period): Participants (par) aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag for 24 weeks. The starting dose for Cohort 1 was 25 mg, and par of East Asian ancestry received 12.5mg QD. For cohort 2 starting dose was based on the body weight. Par with a bodyweight of <27 kg received 12.5 mg QD, par with a body weight of >=27 kg received 25 mg QD; par of east Asian ancestry with a body weight <27 kg received 12.5 mg QD, and with a body weight of >=27 kg received 25 mg QD. For Cohort 3, the starting dose was 0.7 mg/kg QD and 0.5 mg/kg/day for par of East Asian ancestry and the dose calculations were based on the body weight. The maximum dose allowed for all Cohorts was 75mg daily. For all par, individual dose titration was allowed based upon platelet response.
- Part 2/ 3 (Eltrombopag Open-Label Period): Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3: 1 to 5 years), completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet or dry powder for oral suspension in Part 2/3. Par who received eltrombopag during the Randomized Period continued on the same dose, unless adjustments were warranted according to the dosing guidelines, for 17 additional weeks (for a total of 24 weeks of treatment). Par who received placebo during the Randomized Period followed the starting doses for each age Cohort specified for Part 2, and received a total of 24 weeks of eltrombopag treatment.
Arm/Group | Part 1 (Dose-Finding Period) | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag | Part 2/ 3 (Eltrombopag Open-Label Period)
Number analyzed (Participants) | 15 | 21 | 44 | 65
Participants
  Erythrocytes high, n=15, 21, 44, 65 | 5 | 0 | 7 | 15
  Erythrocytes low, n=15, 21, 44, 65 | 2 | 8 | 13 | 24
  Hemoglobin, high, n= 15, 21, 44, 65 | 2 | 2 | 2 | 8
  Hemoglobin low, n= 15, 21, 44, 65 | 10 | 5 | 15 | 32
  Hematocrit, high, n=15, 21, 44, 65 | 1 | 0 | 0 | 5
  Hematocrit, low, n=15, 21, 44, 65 | 10 | 11 | 22 | 39
  Platelets, high, n=15, 21, 44, 65 | 9 | 0 | 6 | 14
  Platelets, low, n=15, 21, 44, 65 | 15 | 21 | 44 | 65
  Leukocytes, high, n=15, 21, 44, 65 | 6 | 5 | 8 | 27
  Leukocytes, low, n=15, 21, 44, 65 | 4 | 5 | 10 | 19
  Neutrophils, high, n=15, 21, 44, 65 | 7 | 5 | 11 | 33
  Neutrophils, low, n=15, 21, 44, 65 | 3 | 4 | 10 | 21
  Lymphocytes, high, n=15, 21, 44, 65 | 1 | 3 | 5 | 11
  Lymphocytes, low, n=15, 21, 44, 65 | 5 | 6 | 10 | 25
  Monocytes, high, n=15, 21, 44, 65 | 3 | 3 | 7 | 15
  Monocytes, low, n=15, 21, 44, 65 | 4 | 7 | 10 | 23
  Eosinophils, high, n=15, 21, 44, 65 | 5 | 3 | 11 | 24
  Eosinophils, low, n=15, 21, 44, 65 | 4 | 2 | 5 | 9
  Basophils, high, n=15, 21, 44, 65 | 6 | 5 | 10 | 20
  Basophils, low, n=15, 21, 44, 65 | 2 | 0 | 1 | 1
  Mean Platelet Volume, high, n=12, 17, 40, 59 | 10 | 10 | 23 | 47
  Mean Platelet Volume, low, n=12, 17, 40, 59 | 4 | 6 | 10 | 16

22. Secondary Outcome: Number of Participants With the Indicated Renal Parameters Falling Outside of the Reference Range Any Time Post-Baseline During Part 1, Part 2, and Part 2/3
Description: Renal parameters included: creatinine (RR: 44.2 - 88.4 umol/L), creatinine clearance derived (RR: 89.0 - 165.0 milliliter per minute [ ml/min]), protein/creatinine (RR: 0.113- 18.0992 microgram per millimoles [mg/mmol]), and urea (RR: 1.785- 8.925 mmol/L). Baseline values were obtained at Day 1. The number of participants with the indicated renal parameters data outside the reference range (with high and low) any time post-Baseline are presented. Anytime post-Baseline assesments included any scheduled and unscheduled post-baseline assessment
Time Frame: Post-Baseline from Week 1 through Follow-up up to Study Week 35
Population: as for outcome 20
Measure: Number; unit: Participants
Groups:
- Part 1 (Dose-Finding Period): Participants aged between 1 and 17 years (Cohort 1 age group- 12 to 17 years, Cohort 2- 6 to 11 years and Cohort 3-1 to 5 years) received eltrombopag for 24 weeks. The starting dose for cohort 1 was eltrombopag 25 mg, (East Asian ancestry: 12.5mg, QD). For cohort 2 starting dose was based on the body weight (Weight <27 kg: 25 mg QD, Weight >=27 kg: 50 mg QD; east Asian ancestry subjects Weight <27 kg: 12.5 mg QD, Weight >=27 kg: 25 mg QD). For cohort 1 and 2 maximum dose allowed was 75mg. For cohort 3 starting dose was 0.7 mg/kg, QD and the dose calculations were based on the body weight. For all participants individual dose titration was allowed based upon platelet response.
- Part 2 (Randomized Period) -Placebo: Participants aged between 1 and 17 years (Cohort 1 age group- 12 to 17 years, Cohort 2- 6 to 11 years and Cohort 3- 1 to 5 years) received eltrombopag matching placebo for 7 weeks.
- Part 2 (Randomized Period) - Eltrombopag: Participants aged between 1 and 17 years (Cohort 1 age group- 12 to 17 years, Cohort 2- 6 to 11 years and Cohort 3-1 to 5 years) received eltrombopag for 7 weeks. The starting dose for cohort 1 was eltrombopag 25 mg, (East Asian ancestry: 12.5mg, QD). For cohort 2 starting dose was based on the body weight (Weight <27 kg: 25 mg QD, Weight >=27 kg: 50 mg QD; east Asian ancestry subjects Weight <27 kg: 12.5 mg QD, Weight >=27 kg: 25 mg QD). For cohort 1 and 2 maximum dose allowed was 75mg. For cohort 3 starting dose was 0.7 mg/kg, QD and the dose calculations were based on the body weight. For all participants individual dose titration was allowed based upon platelet response.
Arm/Group | Part 1 (Dose-Finding Period) | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag | Part 2/ 3 (Eltrombopag Open-Label Period)
Number analyzed (Participants) | 15 | 21 | 44 | 65
Participants
  Creatinine, high, n=15, 21, 44, 65 | 1 | 3 | 6 | 13
  Creatinine, low, n=15, 21, 44, 65 | 5 | 4 | 4 | 12
  Creatinine Clearance Derived, high, n=15, 21,44,65 | 11 | 17 | 28 | 46
  Creatinine Clearance Derived, low, n=15, 21,44,65 | 0 | 2 | 3 | 4
  Protein/Creatinine, high, n=12, 19, 38, 58 | 1 | 2 | 4 | 18
  Protein/Creatinine, low, n=12, 19, 38, 58 | 1 | 0 | 0 | 0
  Urea, high, n=15, 21, 44, 65 | 1 | 2 | 2 | 5
  Urea, low, n=15, 21, 44, 65 | 5 | 1 | 9 | 11

23. Secondary Outcome: Number of Participants With a Positive Urine Microscopy Parameters Any Time Post-Baseline During Part 1
Description: Urine microscopy included Red Blood Cell (RBC) casts, white blood cell (WBC) casts, and epithelial renal tubular cell casts. Urine microscopy data was reviewed by the Medical Monitor in order to classify the results as positive or negative. The number of participants with a positive result at any time post Baseline were reported. A positive result indicated if the result was positive for at least one of RBC casts, WBC casts, or epithelial renal tubular cell casts.
Time Frame: From Baseline up to Study Week 24 of Part 1
Population: Safety Population, only those participants enrolled during Part 1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Epithelial Renal Cell Casts | 0 | 0 | 2
  RBC Casts | 0 | 0 | 0
  WBC Casts | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With a Positive Urine Microscopy Parameters Any Time Post-Baseline During Part 2
Description: Urine microscopy included Red Blood Cell (RBC) casts, white blood cell (WBC) casts, and epithelial renal tubular cell casts. Urine microscopy data was reviewed by the Medical Monitor in order to classify the results as positive or negative. The nmber of participants with positive finding at Baseline and at anytime post-Baseline (Post-BL) were reported. Baseline was defined as the value obtained at the first visit before treatment (Pre-trt). A positive result indicated if the result was positive for at least one of RBC casts, WBC casts, or epithelial renal tubular cell casts.
Time Frame: From Baseline and post-Baseline up to Study Week 7 of Part 2
Population: Safety Population, only those participants enrolled during Part 2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 17 | 4 | 11
Participants
  Pre-trt Epithelial Renal Tubular Cell Casts | 0 | 2 | 0 | 0 | 0 | 0
  Pre-trt RBC Casts | 0 | 1 | 0 | 0 | 0 | 0
  Pre-trt WBC Casts | 0 | 0 | 0 | 0 | 0 | 0
  Post-BL Epithelial Renal Tubular Cell Casts | 1 | 3 | 0 | 0 | 1 | 0
  Post-BL RBC Casts | 0 | 0 | 0 | 0 | 0 | 0
  Post-BL WBC Casts | 0 | 0 | 0 | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With a Positive Urine Microscopy Parameters Any Time Post-Baseline During Part 2/3
Description: Urine microscopy included Red Blood Cell (RBC) casts, white blood cell (WBC) casts, and epithelial renal tubular cell casts. Urine microscopy data was reviewed by the Medical Monitor in order to classify the results as positive or negative. The number of participants with positive finding at Baseline and at anytime post-Baseline (Post-BL) were reported. Baseline was defined as the value obtained at the first visit before treatment (Pre-trt). A positive result indicated if the result was positive for at least one of RBC casts, WBC casts, or epithelial renal tubular cell casts. Participants randomized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: From Baseline and post-Baseline up to Study Week 31 of Part 2/3
Population: Safety Population, only those participants enrolled during Part 2/3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Participants
  Pre-trt Epithelial Renal Tubular Cell Casts | 3 | 0 | 1
  Pre-trt RBC Casts | 1 | 0 | 0
  Pre-trt WBC Casts | 0 | 0 | 0
  Post-BL Epithelial Renal Tubular Cell Casts | 3 | 2 | 1
  Post-BL RBC Casts | 0 | 0 | 1
  Post-BL WBC Casts | 1 | 0 | 1

26. Secondary Outcome: Number of Participants With the Indicated Vital Signs Falling Outside of the Reference Range During Part 1, Part 2, and Part 2/3
Description: Vital sign assessments included systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurements that were measured before any blood draw at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, at each Follow-up week (Week 1-4) and the maximum post- Baseline (BL) visit. BL is defined as the value obtained on Day 1of treatment. The maximum post-BL visit (MPB) included any scheduled and unscheduled post-BL assessment. Reference ranges (RR) for SBP (mmHg) (Lower limit of normal, normal, Upper limit of normal) for Cohort 1: <85, 85-115, >115; for Cohort 2: <85, 85-120,>120; and Cohort 3: <95, 95-135, >135. RR for DBP (mmHg) for Cohort 1: <45, 45-70,>70; for Cohort 2: <50, 50-75, >75; and Cohort 3: <55, 55-85, >85.
Time Frame: From Baseline through Study Week 35
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Groups:
- Part 2 Randomized Period - Placebo: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag matching placebo for 7 weeks.
- Part 2 Randomized Period - Eltrombopag: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag for 7 weeks. The starting dose for Cohort 1 was 37.5 mg QD. For Cohort 2, starting dose was based on the body weight. Par with a body weight of <27 kg received 25 mg QD, and par with a body weight of >=27 kg received 50 mg QD. Par of East Asian ancestry with a body weight of <27 kg received 12.5 mg QD, and with a body weight of >=27 kg received 25 mg QD. For Cohort 3, the starting dose was 1.5 mg/kg QD and 0.8 mg/kg/day for par of East Asian ancestry. The maximum dose allowed was 2mg/kg and could not exceed 75 mg daily. For all par, individual dose titration was allowed based upon platelet response.
Arm/Group | Part 1 Eltrombopag Dose-Finding Period | Part 2 Randomized Period - Placebo | Part 2 Randomized Period - Eltrombopag | Part 2/ 3 (Eltrombopag Open-Label Period)
Number analyzed (Participants) | 15 | 21 | 44 | 65
Participants
  Screening, DBP, high, n=15 ,20 ,41 ,40 | 1 | 4 | 3 | 3
  Screening, DBP, low, n=15, 20, 41, 40 | 0 | 2 | 6 | 5
  Day 1, DBP, high, n=14, 18, 38, 59 | 2 | 4 | 3 | 7
  Day 1, DBP, low, n=14, 18, 38, 59 | 1 | 1 | 3 | 4
  Week 1, DBP, high, n=14, 19, 42, 63 | 1 | 3 | 4 | 5
  Week 1, DBP, low, n=14, 19, 42, 63 | 1 | 1 | 4 | 5
  Week 2, DBP, high, n=15, 20, 42, 61 | 3 | 2 | 2 | 3
  Week 2, DBP, low, n=15, 20, 42, 61 | 2 | 3 | 4 | 5
  Week 3, DBP, high,n=15, 21, 41, 60 | 1 | 3 | 3 | 6
  Week 3, DBP, low,n=15, 21, 41, 60 | 2 | 3 | 5 | 5
  Week 4, DBP,high, n=15, 21, 42, 62 | 0 | 3 | 3 | 6
  Week 4, DBP,low, n=15, 21, 42, 62 | 4 | 4 | 3 | 5
  Week 5, DBP, high, n=15, 19, 40, 59 | 1 | 2 | 4 | 8
  Week 5, DBP, low, n=15, 19, 40, 59 | 1 | 1 | 5 | 5
  Week 6, DBP, high, n=14, 21, 42, 58 | 1 | 2 | 3 | 5
  Week 6, DBP, low, n=14, 21, 42, 58 | 0 | 0 | 3 | 4
  Week 7, DBP, high, n=15, 21, 42, 58 | 1 | 4 | 6 | 7
  Week 7, DBP, low, n=15, 21, 42, 58 | 0 | 1 | 2 | 4
  Week 8, DBP,high,n=15, 0, 0, 49 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  Week 8, DBP,low,n=15, 0, 0, 49 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 6
  Week 9, DBP, high, n=15, 0, 0, 45 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  Week 9, DBP, low, n=15, 0, 0, 45 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 6
  Week 10, DBP, high, n=15, 0, 0, 40 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 6
  Week 10, DBP, low, n=15, 0, 0, 40 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 11, DBP, high, n=13, 0, 0, 41 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  Week 11, DBP, low, n=13, 0, 0, 41 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 12, DBP, high, n=13, 0, 0, 42 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 5
  Week 12, DBP, low, n=13, 0, 0, 42 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 13, DBP, high, n=12, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 13, DBP, low, n=12, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 5
  Week 14, DBP, high, n=9, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 14, DBP, low, n=9, 0, 0, 32 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 15, DBP, high, n=11, 0, 0, 31 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 15, DBP, low, n=11, 0, 0, 31 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 16, DBP,high,n=12, 0, 0, 39 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 16, DBP,low,n=12, 0, 0, 39 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 17, DBP,high,n=5, 0, 0, 29 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 17, DBP,low,n=5, 0, 0, 29 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 18, DBP,high,n=9, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 18, DBP,low,n=9, 0, 0, 32 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 19, DBP,high,n=5, 0, 0, 34 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 19, DBP,low,n=5, 0, 0, 34 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 20, DBP,high,n=13, 0, 0, 33 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 20, DBP,low,n=13, 0, 0, 33 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 21, DBP,high,n=10, 0, 0, 17 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 21, DBP,low,n=10, 0, 0, 17 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 22, DBP,high,n=11, 0, 0, 23 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 22, DBP,low,n=11, 0, 0, 23 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 23, DBP,high,n=11, 0, 0, 21 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 23, DBP,low,n=11, 0, 0, 21 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 24 DBP,high,n=15, 0, 0, 58 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 5
  Week 24, DBP,low,n=15, 0, 0, 58 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  FU Week 1, DBP,high,n=5, 0, 0, 13 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  FU Week 1, DBP,low,n=5, 0, 0, 13 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  FU Week 2, DBP,high,n=5, 0, 0, 21 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  FU Week 2, DBP,low,n=5, 0, 0, 21 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  FU Week 3, DBP,high,n=5, 0, 0, 14 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  FU Week 3, DBP,low,n=5, 0, 0, 14 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  FU Week 4, DBP,high,n=3, 0, 0, 31 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 7
  FU Week 4, DBP,low,n=3, 0, 0, 31 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 5
  Screening, SBP, high, n=15, 20, 41, 40 | 4 | 4 | 10 | 10
  Screening, SBP, low, n=15, 20, 41, 40 | 3 | 0 | 3 | 2
  Day 1, SBP,high,n=14, 18, 38, 59 | 4 | 5 | 9 | 14
  Day 1, SBP,low,n=14, 18, 38, 59 | 0 | 1 | 4 | 4
  Week 1, SBP,high,n=14, 19, 42, 63 | 3 | 6 | 14 | 18
  Week 1, SBP,low,n=14, 19, 42, 63 | 2 | 0 | 4 | 8
  Week 2, SBP,high,n=15, 20, 43, 62 | 4 | 7 | 7 | 15
  Week 2, SBP,low,n=15, 20, 43, 62 | 1 | 2 | 5 | 6
  Week 3, SBP,high,n=15, 21, 41, 60 | 3 | 4 | 12 | 17
  Week 3, SBP,low,n=15, 21, 41, 60 | 1 | 2 | 2 | 3
  Week 4, SBP,high,n=15, 21, 42, 62 | 4 | 6 | 10 | 16
  Week 4, SBP,low,n=15, 21, 42, 62 | 4 | 1 | 3 | 2
  Week 5, SBP,high,n=15, 19, 40, 59 | 5 | 5 | 13 | 17
  Week 5, SBP, low, n=15, 19, 40, 59 | 2 | 1 | 3 | 3
  Week 6, SBP,high,n=14, 21, 42, 58 | 4 | 8 | 11 | 16
  Week 6, SBP,low,n=14, 21, 42, 58 | 2 | 1 | 3 | 5
  Week 7, SBP,high,n=15, 21, 42, 58 | 5 | 5 | 9 | 13
  Week 7, SBP,low,n=15, 21, 42, 58 | 1 | 0 | 2 | 5
  Week 8, SBP,high,n=15, 0, 0, 49 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 16
  Week 8, SBP,low,n=15, 0, 0, 49 | 4 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  Week 9, SBP,high,n=15, 0, 0, 45 | 4 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 15
  Week 9, SBP,low,n=15, 0, 0, 45 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 10, SBP,high,n=15, 0, 0, 40 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  Week 10, SBP,low,n=15, 0, 0, 40 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 11, SBP,high,n=13, 0, 0, 41 | 4 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 9
  Week 11, SBP,low,n=13, 0, 0, 41 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 12, SBP,high,n=13, 0, 0, 42 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  Week 12, SBP,low,n=13, 0, 0, 42 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 13, SBP,high,n=12, 0, 0, 32 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 8
  Week 13, SBP,low,n=12, 0, 0, 32 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 14, SBP,high,n=9, 0, 0, 32 | 4 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  Week 14, SBP,low,n=9, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  Week 15, SBP,high,n=11, 0, 0, 31 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 9
  Week 15, SBP,low,n=11, 0, 0, 31 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 16 SBP,high,n=12, 0, 0, 39 | 5 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 14
  Week 16, SBP,low,n=12, 0, 0, 39 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 17, SBP,high,n=5, 0, 0, 29 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 9
  Week 17, SBP,low,n=5, 0, 0, 29 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 18, SBP,high,n=9, 0, 0, 32 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  Week 18, SBP,low,n=9, 0, 0, 32 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 19, SBP,high,n=5, 0, 0, 34 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 9
  Week 19, SBP,low,n=5, 0, 0, 34 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  Week 20, SBP,high,n=13, 0, 0, 33 | 6 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  Week 20, SBP,low,n=13, 0, 0, 33 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 21, SBP,high,n=10, 0, 0, 17 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 21, SBP,low,n=10, 0, 0, 17 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 22, SBP,high,n=11, 0, 0, 23 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 8
  Week 22, SBP,low,n=11, 0, 0, 23 | 3 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  Week 23, SBP,high,n=11, 0, 0, 21 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 6
  Week 23, SBP,low,n=11, 0, 0, 21 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 1
  Week 24, SBP,high,n=15, 0, 0, 58 | 4 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 19
  Week 24, SBP, low, n=15, 0, 0, 58 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 2
  FU Week 1, SBP, high,n=5, 0, 0, 13 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  FU Week 1, SBP, low,n=5, 0, 0, 13 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  FU Week 2, SBP, high,n=5, 0, 0, 21 | 2 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  FU Week 2, SBP, low,n=5, 0, 0, 21 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3
  FU Week 3, SBP, high,n=5, 0, 0, 14 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 4
  FU Week 3, SBP, low,n=5, 0, 0, 14 | 0 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 0
  FU Week 4, SBP, high,n=3, 0, 0, 31 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 10
  FU Week 4, SBP,low,n=3, 0, 0, 31 | 1 | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | NA — Part 2 ended at Week 7 so no participants were analyzed for this parameter at this time point. | 3

27. Secondary Outcome: Mean Respiratory Rate at Baseline and the Maximum Post-Baseline Value Recorded During the Dose-Finding Period, Part 1
Description: Respiratory rate was measured at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, and at each Follow-up Weeks 1-4. Baseline is defined as the value obtained on Day 1 of treatment. The maximum post-Baseline value included any scheduled and unscheduled post-Baseline assessment.
Time Frame: From Baseline through Week 24
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population .
Measure: Mean (Standard Deviation); unit: Breaths per min
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Breaths per min
  BL, n=4, 5, 4 | 20.0 (0.00) | 21.4 (4.10) | 25.5 (4.43)
  Week 1, n=4,5,4 | 21.5 (4.43) | 22.0 (6.00) | 26.5 (6.40)
  Week 2, n=5,5,4 | 20.6 (3.44) | 19.4 (4.98) | 24.0 (5.42)
  Week 3, n=5,5,5 | 22.0 (5.66) | 17.0 (5.10) | 23.6 (6.07)
  Week 4, n=5,5,5 | 18.8 (1.79) | 17.2 (4.82) | 25.4 (5.98)
  Week 5, n=5,5,4 | 20.4 (2.19) | 20.2 (6.87) | 24.3 (5.56)
  Week 6, n=5,5,4 | 18.4 (2.61) | 20.2 (5.02) | 24.5 (2.52)
  Week 7, n=5,5,5 | 19.2 (1.10) | 23.4 (9.15) | 24.4 (6.69)
  Week 8, n=5,5,5 | 19.8 (3.03) | 20.4 (3.05) | 23.8 (4.82)
  Week 9, n=5,4,5 | 19.2 (2.28) | 22.5 (3.79) | 22.0 (2.00)
  Week 10, n=5,5,5 | 19.6 (2.61) | 18.0 (4.00) | 22.4 (1.67)
  Week 11, n=5,3,4 | 19.6 (1.67) | 20.3 (3.21) | 25.0 (5.03)
  Week 12, n=4,3,4 | 19.5 (1.00) | 20.0 (0.00) | 27.6 (11.52)
  Week 13, n=4,4,4 | 19.5 (1.00) | 21.0 (2.16) | 23.0 (3.46)
  Week 14, n=3,3,3 | 18.7 (1.15) | 22.7 (1.15) | 27.3 (7.57)
  Week 15, n=3,3,3 | 18.0 (2.00) | 21.3 (1.15) | 24.0 (2.00)
  Week 16, n=5,3,4 | 18.8 (3.35) | 20.0 (4.00) | 30.8 (16.88)
  Week 17, n=2,0,3 | 18.0 (0.00) | NA (NA) — No participants were analyzed for this parameter at this time point. | 24.0 (4.00)
  Week 18, n=3,3,4 | 19.3 (1.15) | 21.3 (3.06) | 29.0 (13.22)
  Week 19, n=3,0,2 | 19.3 (1.15) | NA (NA) — No participants were analyzed for this parameter at this time point. | 28.0 (11.31)
  Week 20, n=5,4,4 | 19.6 (1.67) | 21.5 (3.00) | 23.5 (3.42)
  Week 21, n=3,2,5 | 19.3 (1.15) | 19.00 (1.41) | 23.6 (3.51)
  Week 22, n=3,4,3 | 19.3 (2.31) | 21.0 (2.00) | 27.3 (7.57)
  Week 23, n=4,2,4 | 20.0 (1.63) | 20.0 (0.00) | 21.5 (1.91)
  Week 24, n=5,5,4 | 19.6 (0.89) | 23.0 (3.16) | 24.8 (7.09)
  FU Week 1, n=1,1,3 | 20.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 20.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 22.0 (2.00)
  FU Week 2, n=3,2,0 | 19.3 (1.15) | 26.5 (9.19) | NA (NA) — No participants were analyzed for this parameter at this time point.
  FU Week 3, n=2,1,2 | 21.0 (4.24) | 28.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 24.5 (4.95)
  FU Week 4, n=1,0,1 | 18.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | NA (NA) — No participants were analyzed for this parameter at this time point. | 24.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation.
  MPB, n=5, 5, 5 | 24.4 (4.56) | 29.8 (6.02) | 32.2 (13.90)

28. Secondary Outcome: Mean Respiratory Rate at Baseline and the Maximum Post-Baseline Value Recorded During the Randomized Period, Part 2
Description: as for outcome 27
Time Frame: From Week 1 to Week 7 of Part 2
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X,X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety Population
Measure: Mean (Standard Deviation); unit: Breaths per min
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 17 | 4 | 11
Breaths per min
  BL, n= 5, 14, 9, 12, 3, 10 | 19.6 (1.67) | 18.4 (2.38) | 19.4 (3.13) | 21.5 (10.03) | 18.7 (1.15) | 21.4 (2.12)
  Week 1, n=7, 16 ,9, 17, 2, 10 | 19.0 (1.00) | 18.8 (1.76) | 19.9 (2.26) | 20.7 (4.48) | 19.0 (1.41) | 28.2 (9.54)
  Week 2, n=6, 15, 9, 16, 4, 10 | 19.3 (2.73) | 18.9 (2.70) | 19.8 (2.33) | 23.0 (8.01) | 21.5 (5.00) | 27.1 (11.70)
  Week 3, n=8, 16, 9, 16, 4, 9 | 18.8 (1.83) | 18.9 (1.93) | 20.1 (2.76) | 22.3 (4.78) | 21.0 (2.58) | 25.8 (7.17)
  Week 4, n=7, 16, 8, 14, 4, 10 | 19.4 (2.51) | 18.6 (2.80) | 19.8 (2.49) | 21.4 (4.29) | 21.5 (1.00) | 25.4 (7.18)
  Week 5, n=8, 16, 8, 15, 3, 8 | 19.3 (1.04) | 18.5 (2.10) | 20.5 (2.98) | 19.7 (2.74) | 20.0 (2.00) | 29.0 (14.77)
  Week 6, n=8, 16, 9, 15, 4, 9 | 20.3 (2.25) | 19.4 (2.16) | 20.6 (2.19) | 20.6 (4.12) | 21.0 (1.15) | 24.4 (6.69)
  Week 7, n=7, 16, 9, 17, 4, 8 | 20.9 (2.27) | 18.4 (1.50) | 20.9 (3.33) | 20.7 (7.87) | 18.5 (1.91) | 23.5 (6.12)
  MPB, n=8, 16, 9, 17, 4, 11 | 21.5 (2.33) | 21.3 (21.8) | 22.7 (2.45) | 26.6 (7.87) | 23.5 (3.42) | 30.0 (13.39)

29. Secondary Outcome: Mean Respiratory Rate at Baseline and Maximum Post-Baseline Visit During Part 2/3
Description: Respiratory rate was measured at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, and at each Follow-up Weeks 1-4. Baseline is defined as the value obtained on Day 1 of treatment. The maximum post-Baseline visit included any scheduled and unscheduled post-Baseline assessment. Participants randomized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: From Week 1 to Follow-up Week 4 of Part 2/3 up to Study Week 35
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2/3 (Eltrombopag Period) Cohort 1 | Part 2/3 (Eltrombopag Period) Cohort 2 | Part 2/3 (Eltrombopag Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Breaths per minute
  Screening, n=16, 14, 10 | 18.5 (1.75) | 21.2 (6.57) | 21.5 (2.56)
  Day 1 , n=21, 21, 15 | 19.2 (2.57) | 2.12 (7.74) | 21.7 (4.76)
  Week 1, n=24, 25, 14 | 19.1 (1.74) | 20.4 (3.93) | 25.1 (7.63)
  Week 2, n=22, 24, 13 | 19.4 (2.56) | 21.8 (6.85) | 25.2 (10.83)
  Week 3, n=24, 23, 12 | 18.8 (1.73) | 21.2 (4.40) | 24.0 (6.09)
  Week 4, n=23, 23, 13 | 19.0 (2.59) | 20.9 (3.82) | 24.3 (6.37)
  Week 5, n=23, 23, 11 | 18.9 (2.13) | 19.8 (3.19) | 26.9 (12.91)
  Week 6, n=23, 22, 11 | 19.3 (2.30) | 20.6 (4.11) | 23.3 (4.92)
  Week 7, n=22, 25, 11 | 18.8 (1.99) | 20.1 (4.46) | 22.4 (4.60)
  Week 8, n=19, 19, 10 | 19.2 (2.32) | 23.4 (6.23) | 22.0 (1.79)
  Week 9, n=17, 16, 12 | 19.5 (2.96) | 22.0 (3.95) | 22.5 (4.48)
  Week 10, n=16, 13, 11 | 18.7 (2.27) | 22.8 (3.83) | 23.3 (6.83)
  Week 11, n=15, 13, 12 | 18.9 (1.28) | 22.8 (3.11) | 22.2 (5.29)
  Week 12, n=17, 16, 9 | 18.6 (1.90) | 22.2 (3.76) | 23.6 (4.98)
  Week 13, n=11, 13, 8 | 19.3 (1.56) | 23.4 (7.68) | 21.0 (2.62)
  Week 14, n=13, 11, 7 | 18.7 (2.98) | 19.9 (5.49) | 23.4 (4.86)
  Week 15, n=12, 13, 5 | 18.7 (1.76) | 21.1 (2.53) | 24.4 (8.76)
  Week 16, n=16, 14, 8 | 18.6 (1.26) | 22.9 (7.97) | 24.3 (6.88)
  Week 17, n=13, 10, 5 | 19.0 (2.08) | 22.4 (6.45) | 25.2 (9.65)
  Week 18, n=16, 12, 4 | 19.1 (3.79) | 22.0 (4.53) | 29.0 (10.52)
  Week 19, n=14, 13, 6 | 18.1 (1.49) | 24.5 (19.33) | 24.0 (6.45)
  Week 20, n=13, 13, 7 | 17.4 (1.94) | 20.9 (3.52) | 33.00 (16.77)
  Week 21, n=4, 10, 3 | 18.8 (3.40) | 20.2 (3.55) | 28.0 (10.58)
  Week 22, n=11, 7, 5 | 19.7 (2.94) | 19.1 (2.79) | 26.0 (4.90)
  Week 23, n=8, 7, 6 | 20.4 (2.72) | 21.1 (3.24) | 23.7 (5.13)
  Week 24, n=22, 23, 11 | 19.1 (2.03) | 20.2 (3.11) | 23.8 (5.47)
  FU Week 1, n=6, 6, 3 | 18.8 (1.60) | 20.0 (3.41) | 26.0 (10.39)
  FU Week 2, n=6, 5, 7 | 18.7 (1.63) | 20.8 (4.15) | 22.2 (4.02)
  FU Week 3, n=6, 4, 4 | 19.0 (1.67) | 23.0 (4.16) | 24.8 (5.50)
  FU Week 4, n=10, 12, 7 | 19.4 (0.97) | 20.8 (1.86) | 21.0 (3.74)
  MPB, n=24, 26, 15 | 23.0 (2.78) | 27.7 (13.00) | 27.7 (11.54)

30. Secondary Outcome: Mean Pulse Rate at Baseline and the Maximum Post-Baseline Visit Recorded During the Dose-Finding Period, Part 1
Description: Pulse rate was measured at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, and at each Follow-up Weeks 1-4. Baseline is defined as the value obtained on Day 1 of treatment. The maximum post-Baseline (MPB) visit included any scheduled and unscheduled post-Baseline assessment..
Time Frame: From Week 1 to Follow-up Week 4 of Part 1, up to Study Week 28
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Beats per minute
  Screening, n=5, 5, 5 | 85.2 (15.71) | 88.4 (8.50) | 102.0 (7.97)
  Day 1, n=4, 5, 5, | 84.3 (11.32) | 88.2 (12.89) | 102.4 (13.22)
  Week 1, n= 4, 5, 5 | 85.3 (4.79) | 90.8 (11.19) | 103.8 (8.47)
  Week 2, n=5, 5, 5 | 80.4 (12.97) | 84.4 (16.77) | 96.8 (10.66)
  Week 3, n=5, 5, 5 | 92.8 (31.16) | 91.4 (11.04) | 106.2 (11.10)
  Week 4, n=5, 5, 5 | 86.4 (10.92) | 84.0 (7.62) | 98.6 (14.29)
  Week 5, n=5, 5, 5 | 84.6 (9.48) | 88.4 (9.58) | 107.8 (9.58)
  Week 6, n=5, 5, 4 | 76.4 (10.50) | 89.8 (13.79) | 103.0 (8.29)
  Week 7, n=5, 5, 5 | 82.0 (9.46) | 96.2 (17.84) | 103.2 (8.93)
  Week 8, n=5, 5, 5 | 83.0 (5.20) | 89.4 (15.04) | 111.8 (10.62)
  Week 9, n=5, 5, 5 | 80.4 (13.35) | 79.2 (11.34) | 101.6 (5.59)
  Week 10, n=5, 5, 5 | 80.6 (14.93) | 84.4 (10.31) | 105.4 (9.29)
  Week 11, n=5, 3, 5 | 86.6 (11.04) | 97.7 (16.50) | 106.6 (11.19)
  Week 12, n=4, 4, 5 | 80.5 (12.07) | 92.0 (12.83) | 101.4 (16.62)
  Week 13, n=4, 4, 4 | 90.8 (15.52) | 86.5 (7.05) | 103.8 (3.50)
  Week 14, n=3, 3, 3 | 81.0 (9.85) | 87.0 (8.66) | 101.0 (11.00)
  Week 15, n=3, 4, 4 | 77.3 (6.66) | 86.8 (11.87) | 102.5 (3.87)
  Week 16, n=5, 3, 4 | 86.4 (18.60) | 103.0 (5.57) | 93.0 (18.96)
  Week 17, n=2, 0, 3 | 67.5 (20.51) | NA (NA) — There were no participants analyzed at this time point, therefore there is no calculated standard deviation. | 97.7 (12.01)
  Week 18, n=3, 3, 4 | 88.0 (10.44) | 86.7 (17.01) | 102.8 (16.88)
  Week 19, n=3, 0, 2 | 88.0 (20.81) | NA (NA) — There were no participants analyzed at this time point, therefore there is no calculated standard deviation. | 94.0 (8.49)
  Week 20, n=5, 4, 4 | 79.8 (13.03) | 96.8 (12.58) | 111.8 (14.97)
  Week 21, n=3, 2, 5 | 79.0 (6.93) | 75.5 (3.54) | 101.0 (18.63)
  Week 22, n=3, 4, 4 | 70.3 (14.36) | 86.5 (9.04) | 100.0 (18.63)
  Week 23, n=4, 2, 5 | 71.5 (13.03) | 82.5 (3.54) | 100.0 (13.14)
  Week 24, n=5, 5, 5 | 79.6 (7.86) | 85.8 (6.91) | 96.0 (4.74)
  FU Week 1, n=1, 1, 3 | 81.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 125.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 107.7 (10.79)
  FU Week 2, n=3, 2, 0 | 77.7 (8.74) | 84.5 (28.99) | NA (NA) — There were no participants analyzed at this time point, therefore there is no calculated standard deviation.
  FU Week 3, n=2, 1, 2 | 87.0 (2.83) | 78.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | 98.0 (8.49)
  FU Week 4, n=1, 0, 2 | 89.0 (NA) — There were too few participants available to collect data at this time point to calculate a standard deviation. | NA (NA) — There were no participants analyzed at this time point, therefore there is no calculated standard deviation. | 99.0 (26.87)
  MBP, n=5, 5, 5 | 108.8 (24.01) | 109.8 (14.17) | 119.6 (5.73)

31. Secondary Outcome: Mean Pulse Rate at Baseline and the Maximum Post-Baseline Visit Recorded During the Randomized Period, Part 2
Description: Pulse rate was measured at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, and at each Follow-up Weeks 1-4. Baseline is defined as the value obtained on Day 1 of treatment. The maximum post-Baseline visit included any scheduled and unscheduled post-Baseline assessment.
Time Frame: From Week 1 to Week 7 of Part 2
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X,X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 17 | 4 | 11
Beats per minute
  Screening, n=8, 16, 9, 15 | 80.1 (10.11) | 82.8 (17.28) | 86.9 (16.10) | 94.3 (17.53) | 91.5 (6.56) | 101.5 (23.48)
  Day 1, n=6, 14, 9, 13 | 77.2 (12.32) | 81.3 (8.70) | 93.0 (14.04) | 88.8 (12.84) | 98.7 (5.69) | 99.6 (15.84)
  Week 1, n=8, 16, 9, 17 | 76.4 (8.50) | 80.1 (12.04) | 89.9 (18.48) | 98.4 (19.76) | 98.5 (13.44) | 96.4 (17.08)
  Week 2, n=7, 15, 9, 17 | 79.4 (8.75) | 81.7 (9.79) | 89.0 (12.44) | 91.8 (16.96) | 95.3 (7.09) | 102.5 (11.81)
  Week 3, n=8, 16, 9, 16 | 81.5 (12.21) | 84.0 (10.93) | 86.6 (13.39) | 95.8 (13.57) | 97.0 (14.67) | 102.6 (17.44)
  Week 4, n=8, 16, 9, 16 | 76.3 (6.96) | 82.4 (10.39) | 84.4 (15.91) | 91.5 (14.45) | 93.5 (17.00) | 116.1 (23.26)
  Week 5, n=8, 16, 9, 16 | 79.3 (9.44) | 82.5 (13.87) | 95.3 (14.96) | 92.4 (15.18) | 89.0 (15.52) | 99.8 (19.51)
  Week 6, n=8, 16, 9, 17 | 77.0 (9.50) | 83.2 (11.01) | 86.8 (11.62) | 90.1 (17.74) | 84.8 (13.15) | 103.0 (23.14)
  Week 7, n=8, 16, 9, 17 | 74.1 (6.92) | 82.8 (11.68) | 96.7 (15.39) | 91.6 (17.68) | 101.5 (16.60) | 105.3 (15.18)
  MBP, n=8, 16, 9, 17 | 88.3 (7.72) | 97.6 (7.51) | 106.1 (11.92) | 108.6 (17.08) | 106.8 (12.28) | 117.5 (21.68)

32. Secondary Outcome: Mean Pulse Rate at Baseline and the Maximum Post-Baseline Visit Recorded During the Eltrombopag Only Period Part 2/3
Description: Pulse rate was measured at the following scheduled time points: Screening, Day 1, each week from Week 1 to Week 24, and at each Follow-up Weeks 1-4. Baseline is defined as the value obtained on Day 1 of treatment. The maximum post-Baseline visit included any scheduled and unscheduled post-Baseline assessment. Participants randomized to receive eltrombopag for 7 weeks in Part 2 continued receiving eltrombopag for an additional 17 weeks in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 24. Participants randomized to receive placebo for 7 weeks in Part 2, received 24 weeks of eltrombopag in Part 2/3 (for a total of 24 weeks of treatment) up to Study Week 31.
Time Frame: From Week 1to Follow-up Week 4 of Part 2/3, up to Study Week 35
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2/3 (Eltrombopag Period) Cohort 1 | Part 2/3 (Eltrombopag Period) Cohort 2 | Part 2/3 (Eltrombopag Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Beats per minute
  Screening, n=16, 15, 10 | 82.8 (17.28) | 94.3 (17.53) | 104.8 (21.82)
  Day 1 , n=22, 22, 15 | 78.7 (8.67) | 92.0 (14.14) | 100.8 (15.71)
  Week 1, n=24, 26, 14 | 79.9 (10.82) | 94.8 (17.54) | 97.8 (15.67)
  Week 2, n=23, 26, 13 | 79.9 (10.02) | 92.5 (16.91) | 99.8 (12.64)
  Week 3, n=24, 24, 12 | 83.3 (10.63) | 95.4 (12.31) | 99.4 (16.56)
  Week 4, n=24, 25, 13 | 81.9 (9.81) | 91.7 (13.42) | 110.6 (22.55)
  Week 5, n=24, 24, 11 | 80.8 (13.00) | 91.7 (14.72) | 97.4 (17.92)
  Week 6, n=23, 24, 11 | 82.2 (10.45) | 91.6 (16.82) | 102.8 (20.31)
  Week 7, n=22, 25, 11 | 82.1 (11.47) | 91.1 (16.61) | 101.5 (16.91)
  Week 8, n=19, 20, 10 | 79.9 (11.85) | 90.8 (16.68) | 94.2 (25.71)
  Week 9, n=17, 16, 12 | 87.4 (15.75) | 91.9 (17.79) | 100.9 (15.19)
  Week 10, n=16, 13, 11 | 87.9 (11.74) | 94.3 (17.82) | 97.8 (18.77)
  Week 11, n=15, 14, 12 | 81.5 (10.20) | 89.3 (16.28) | 99.3 (15.39)
  Week 12, n=17, 16, 9 | 81.1 (11.98) | 91.1 (16.39) | 105.3 (19.58)
  Week 13, n=11, 13, 8 | 78.1 (8.47) | 97.0 (21.79) | 99.5 (20.57)
  Week 14, n=13, 12, 7 | 74.5 (11.15) | 94.8 (18.07) | 95.6 (12.09)
  Week 15, n=12, 14, 5 | 82.5 (9.41) | 94.4 (18.94) | 98.0 (8.72)
  Week 16, n=17, 14, 8v | 81.3 (11.24) | 91.4 (15.08) | 99.8 (17.16)
  Week 17, n=13, 11, 5 | 79.7 (11.69) | 96.1 (20.80) | 102.2 (22.61)
  Week 18, n=16, 12, 4 | 81.1 (8.79) | 95.8 (23.01) | 99.8 (5.56)
  Week 19, n=14, 14, 6 | 82.1 (12.33) | 96.5 (20.24) | 104.2 (18.88)
  Week 20, n=13, 13, 7 | 79.0 (10.98) | 95.9 (17.44) | 91.6 (17.18)
  Week 21, n=4, 10, 3 | 82.3 (10.53) | 90.3 (10.71) | 99.7 (15.28)
  Week 22, n=11, 6, 5 | 83.2 (10.57) | 99.7 (5.50) | 98.6 (18.20)
  Week 23, n=8, 7, 6 | 80.4 (11.25) | 89.0 (22.38) | 96.2 (10.68)
  Week 24, n=23, 23, 11 | 81.2 (9.70) | 93.5 (12.59) | 95.3 (17.75)
  FU Week 1, n=6, 6, 3 | 86.3 (5.85) | 94.2 (18.03) | 100.0 (20.07)
  FU Week 2, n=8, 7, 7 | 83.0 (8.54) | 87.9 (12.77) | 110.0 (27.47)
  FU Week 3, n=6, 5, 4 | 83.7 (13.03) | 92.4 (11.55) | 92.0 (12.19)
  FU Week 4, n=11, 13, 7 | 81.6 (11.89) | 92.3 (16.10) | 102.3 (18.87)
  MPB, n=24, 26, 15 | 102.2 (9.35) | 110.9 (15.03) | 121.2 (20.42)

33. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick at Baseline and Week 24 During the Dose-Finding Period, Part 1
Description: Urinalysis parameters included: urine protein (UP), urine glucose (UG), urine ketones (UK), urine occult blood (UOB), and pH. The dipstick test gives results in a semi-quantitative manner. UP was categorized as missing (MS), no result (NR), negative (Neg), Trace, 1+, 2+, 3+ and 4+. UG results were categorized as MS, NR, Neg, normal, 5, 15(1+), 30(2+), 60(3+), 110(4+)UK parameters were categorized as as MS, NR, Neg, Trace(5), Small(15), Moderate(40), Large(80), Large(160). UOB parameters were categorized as MS, NR, Neg, 1+, 2+, 3+, Non haemolysed trace, and haemolysed trace. PH results were categorized as MS. NR, normalresult, Neg, and range of pH (from 5-9in increments of 0.5). Data for indicated parameters was reported at Baseline (BL) and Week 24 (W24). The Baseline value was the measurement taken at Day 1.
Time Frame: Baseline and Week 24 of Part 1
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1 Eltrombopag Dose-Finding Period
Number analyzed (Participants) | 15
Participants
  UP, MS, BL, n=3 | 1
  UP, NR, BL, n=3 | 0
  UP, Neg, BL, n=3 | 0
  UP, Trace, BL, n=3 | 2
  UP, 1+, BL, n=3 | 0
  UP, 2+, BL, n=3 | 0
  UP, 3+, BL, n=3 | 0
  UP, 4+, BL, n=3 | 0
  UG, MS, BL, n=3 | 0
  UG, NR, BL, n=3 | 0
  UG, Neg, BL, n=3 | 3
  UG, normal, BL, n=3 | 0
  UG, 5, BL, n=3 | 0
  UG, 15(1+), BL, n=3 | 0
  UG, 30(2+), BL, n=3 | 0
  UG, 60(3+), BL, n=3 | 0
  UG, 110(4+), BL, n=3 | 0
  UK, MS, BL, n=3 | 0
  UK, NR, BL, n=3 | 0
  UK, Neg, BL, n=3 | 3
  UK, Trace(5), BL, n=3 | 0
  UK, Small(15), BL, n=3 | 0
  UK, Moderate(40), BL, n=3 | 0
  UK, Large(80), BL, n=3 | 0
  UK, Large(160), BL, n=3 | 0
  UOB, MS, BL,n=3 | 1
  UOB, NR, BL,n=3 | 0
  UOB, Neg, BL,n=3 | 2
  UOB, 1+, BL,n=3 | 0
  UOB, 2+, BL,n=3 | 0
  UOB, 3+, BL,n=3 | 0
  UOB, Non haemolysed trace, BL,n=3 | 0
  UOB, haemolysed trace, BL,n=3 | 0
  pH, MS, BL, n=3 | 0
  pH, NR, BL, n=3 | 0
  pH, normal result, BL, n=3 | 0
  pH, Neg, BL, n=3 | 0
  pH, 5, BL, n=3 | 0
  pH, 5.5, BL, n=3 | 0
  pH, 6, BL, n=3 | 0
  pH, 6.5, BL, n=3 | 1
  pH, 7, BL, n=3 | 0
  pH, 7.5,BL, n=3 | 1
  pH, 8, BL, n=3 | 1
  pH, 8.5, BL, n=3 | 0
  pH, 9, BL, n=3 | 0
  UP, MS, W24, n=4 | 0
  UP, NR, W24, n=4 | 0
  UP, Neg, W24, n=4 | 3
  UP, Trace, W24, n=4 | 1
  UP, 1+, W24, n=4 | 0
  UP, 2+, W24, n=4 | 0
  UP, 3+, W24, n=4 | 0
  UP, 4+, W24, n=4 | 0
  UG, MS, W24, n=4 | 0
  UG, NR, W24, n=4 | 0
  UG, Neg, W24, n=4 | 4
  UG, normal, W24, n=4 | 0
  UG, 5, W24, n=4 | 0
  UG, 15(1+), W24, n=4 | 0
  UG, 30(2+), W24, n=4 | 0
  UG, 60(3+), W24, n=4 | 0
  UG, 110(4+), W24, n=4 | 0
  UK, MS, W24, n=4 | 0
  UK, NR, W24, n=4 | 0
  UK, Neg, W24, n=4 | 3
  UK, Trace(5), W24, n=4 | 1
  UK, Small(15), W24, n=4 | 0
  UK, Moderate(40), W24, n=4 | 0
  UK, Large(80), W24, n=4 | 0
  UK, Large(160), W24, n=4 | 0
  UOB, MS, W24, n=4 | 0
  UOB, NR, W24, n=4 | 0
  UOB, Neg, W24, n=4 | 3
  UOB, 1+, W24, n=4 | 0
  UOB, 2+, W24, n=4 | 0
  UOB, 3+, W24, n=4 | 0
  UOB, Non haemolysed trace, W24, n=4 | 0
  UOB, haemolysed trace, W24, n=4 | 0
  pH, MS, W24, n=4 | 0
  pH, NR, W24, n=4 | 0
  pH, normal result, W24, n=4 | 0
  pH, Neg, W24, n=4 | 0
  pH, 5, W24, n=4 | 0
  pH, 5.5, W24, n=4 | 0
  pH, 6, W24, n=4 | 2
  pH, 6.5, W24, n=4 | 2
  pH, 7, W24, n=4 | 0
  pH, 7.5,W24, n=4 | 0
  pH, 8, W24, n=4 | 0
  pH, 8.5, W24, n=4 | 0
  pH, 9, W24, n=4 | 0

34. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick at Baseline and Week 7 During the Randomized Period,Part 2
Description: Urinalysis parameters included: urine protein (UP), urine glucose (UG), urine ketones (UK), urine occult blood (UOB), and pH. The dipstick test gives results in a semi-quantitative manner. UP was categorized as missing (MS), no result (NR), negative (Neg), Trace, 1+, 2+, 3+ and 4+. UG results were categorized as MS, NR, Neg, normal, 5, 15(1+), 30(2+), 60(3+), 110(4+)UK parameters were categorized as as MS, NR, Neg, Trace(5), Small(15), Moderate(40), Large(80), Large(160). UOB parameters were categorized as MS, NR, Neg, 1+, 2+, 3+, Non haemolysed trace, and haemolysed trace. PH results were categorized as MS. NR, normalresult, Neg, and range of pH (from 5-9in increments of 0.5). Data for indicated parameters was reported at Baseline (BL) and Week 7 (W7). The Baseline value was the measurement taken at Day 1.
Time Frame: Baseline and Week 7 of Part 2
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety Population
Measure: Number; unit: Participants
Groups:
- Part 2 Randomized Period - Placebo: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3:1 to 5 years) received eltrombopag matching placebo QD for 7 weeks.
Arm/Group | Part 2 Randomized Period - Placebo | Part 2 Randomized Period - Eltrombopag
Number analyzed (Participants) | 21 | 44
Participants
  UP, MS, BL, n=10, 9 | 2 | 0
  UP, NR, BL, n=10, 9 | 0 | 1
  UP, Neg, BL, n=10, 9 | 7 | 8
  UP, Trace, BL, n=10, 9 | 1 | 0
  UP, 1+, BL, n=10, 9 | 0 | 0
  UP, 2+, BL, n=10, 9 | 0 | 0
  UP, 3+, BL, n=10, 9 | 0 | 0
  UP, 4+, BL, n=10, 9 | 0 | 0
  UG, MS, BL, n=10, 9 | 2 | 0
  UG, NR, BL, n=10, 9 | 0 | 1
  UG, Neg, BL, n=10, 9 | 6 | 8
  UG, normal, BL, n=10, 9 | 2 | 0
  UG, 5, BL, n=10, 9 | 0 | 0
  UG, 15(1+), BL, n=10, 9 | 0 | 0
  UG, 30(2+), BL, n=10, 9 | 0 | 0
  UG, 60(3+), BL, n=10, 9 | 0 | 0
  UG, 110(4+), BL, n=10, 9 | 0 | 0
  UK, MS, BL, n=10, 9 | 2 | 0
  UK, NR, BL, n=10, 9 | 0 | 1
  UK, Neg, BL, n=10, 9 | 8 | 8
  UK, Trace(5), BL, n=10, 9 | 0 | 0
  UK, Small(15), BL, n=10, 9 | 0 | 0
  UK, Moderate(40), BL, n=10, 9 | 0 | 0
  UK, Large(80), BL, n=10, 9 | 0 | 0
  UK, Large(160), BL, n=10, 9 | 0 | 0
  UOB, MS, BL, n=9, 9 | 2 | 1
  UOB, NR, BL, n=9, 9 | 0 | 1
  UOB, Neg, BL, n=9, 9 | 6 | 4
  UOB, 1+, BL,n=9, 9 | 0 | 1
  UOB, 2+, BL,n=9, 9 | 1 | 0
  UOB, 3+, BL, n=9, 9 | 0 | 0
  UOB, Non haemolysed trace, BL,n=9, 9 | 0 | 0
  UOB, haemolysed trace, BL, n=9, 9 | 0 | 0
  pH, MS, BL, n=10, 9 | 0 | 0
  pH, NR, BL, n=10, 9 | 0 | 1
  pH, normal result, BL, n=10, 9 | 0 | 0
  pH, Neg, BL, n=10, 9 | 0 | 0
  pH, 5, BL, n=10, 9 | 1 | 1
  pH, 5.5, BL, n=10, 9 | 1 | 1
  pH, 6, BL, n=10, 9 | 3 | 4
  pH, 6.5, BL, n=10, 9 | 2 | 1
  pH, 7, BL, n=10, 9 | 1 | 0
  pH, 7.5,BL, n=10, 9 | 1 | 1
  pH, 8, BL, n=10, 9 | 1 | 0
  pH, 8.5, BL, n=10, 9 | 0 | 0
  pH, 9, BL, n=10, 9 | 0 | 0
  UP, MS, W7, n=2, 3 | 0 | 0
  UP, NR, W7, n=2, 3 | 0 | 0
  UP, Neg, W7, n=2, 3 | 2 | 3
  UP, Trace, W7, n=2, 3 | 0 | 0
  UP, 1+, W7, n=2, 3 | 0 | 0
  UP, 2+, W7, n=2, 3 | 0 | 0
  UP, 3+, W7, n=2, 3 | 0 | 0
  UP, 4+, W7, n=2, 3 | 0 | 0
  UG, MS, W7, n=2, 3 | 0 | 0
  UG, NR, W7, n=2, 3 | 0 | 0
  UG, Neg, W7, n=2, 3 | 2 | 3
  UG, normal, W7, n=2, 3 | 0 | 0
  UG, 5, W7, n=2, 3 | 0 | 0
  UG, 15(1+), W7, n=2, 3 | 0 | 0
  UG, 30(2+), W7, n=2, 3 | 0 | 0
  UG, 60(3+), W7, n=2, 3 | 0 | 0
  UG, 110(4+), W7, n=2, 3 | 0 | 0
  UK, MS, W7, n=2, 3 | 0 | 0
  UK, NR, W7, n=2, 3 | 0 | 0
  UK, Neg, W7, n=2, 3 | 2 | 3
  UK, Trace(5), W7, n=2, 3 | 0 | 0
  UK, Small(15), W7, n=2, 3 | 0 | 0
  UK, Moderate(40), W7, n=2, 3 | 0 | 0
  UK, Large(80), W7, n=2, 3 | 0 | 0
  UK, Large(160), W7, n=2, 3 | 0 | 0
  UOB, MS, W7, n=2, 3 | 1 | 0
  UOB, NR, W7, n=2, 3 | 0 | 0
  UOB, Neg, W7, n=2, 3 | 1 | 3
  UOB, 1+, W7, n=2, 3 | 0 | 0
  UOB, 2+, W7, n=2, 3 | 0 | 0
  UOB, 3+, W7, n=2, 3 | 0 | 0
  UOB, Non haemolysed trace, W7, n=2, 3 | 0 | 0
  UOB, haemolysed trace, W7, n=2, 3 | 0 | 0
  pH, MS, W7, n=2, 3 | 0 | 0
  pH, NR, W7, n=2, 3 | 0 | 0
  pH, normal result, W7, n=2, 3 | 0 | 0
  pH, Neg, W7, n=2, 3 | 0 | 0
  pH, 5, W7, n=2, 3 | 1 | 0
  pH, 5.5, W7, n=2, 3 | 0 | 0
  pH, 6, W7, n=2, 3 | 0 | 1
  pH, 6.5, W7, n=2, 3 | 0 | 1
  pH, 7, W7, n=2, 3 | 1 | 1
  pH, 7.5, W7, n=2, 3 | 0 | 0
  pH, 8, W7, n=2, 3 | 0 | 0
  pH, 8.5, W7, n=2, 3 | 0 | 0
  pH, 9, W7, n=2, 3 | 0 | 0

35. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick at Baseline and Week 24 During the Eltrombopag Open-label Period, Part 2/3
Description: as for outcome 33
Time Frame: Baseline and Week 24 of Part 2/3 up to Study Week 31
Population: as for outcome 33
Measure: Number; unit: Participants
Groups:
- Part 2/ 3 Eltrombopag Open-Label Period: Par aged between 1 and 17 years (Cohort 1 age group: 12 to 17 years, Cohort 2: 6 to 11 years and Cohort 3: 1 to 5 years), completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet or dry powder for oral suspension in Part 2/3. Par who received eltrombopag during the Randomized Period continued on the same dose, unless adjustments were warranted according to the dosing guidelines, for 17 additional weeks (for a total of 24 weeks of treatment). Par who received placebo during the Randomized Period followed the starting doses for each age Cohort specified for Part 2, and received a total of 24 weeks of eltrombopag treatment.
Arm/Group | Part 2/ 3 Eltrombopag Open-Label Period
Number analyzed (Participants) | 44
Participants
  UP, MS, BL, n=11 | 0
  UP, NR, BL, n=11 | 1
  UP, Neg, BL, n=11 | 10
  UP, Trace, BL, n=11 | 0
  UP, 1+, BL, n=11 | 0
  UP, 2+, BL, n=11 | 0
  UP, 3+, BL, n=11 | 0
  UP, 4+, BL, n=11 | 0
  UG, MS, BL, n=11 | 0
  UG, NR, BL, n=11 | 1
  UG, Neg, BL, n=11 | 10
  UG, normal, BL, n=11 | 0
  UG, 5, BL, n=11 | 0
  UG, 15(1+), BL, n=11 | 0
  UG, 30(2+), BL, n=11 | 0
  UG, 60(3+), BL, n=11 | 0
  UG, 110(4+), BL, n=11 | 0
  UK, MS, BL, n=11 | 0
  UK, NR, BL, n=11 | 1
  UK, Neg, BL, n=11 | 10
  UK, Trace(5), BL, n=11 | 0
  UK, Small(15), BL, n=11 | 0
  UK, Moderate(40), BL, n=11 | 0
  UK, Large(80), BL, n=11 | 0
  UK, Large(160), BL, n=11 | 0
  UOB, MS, BL,n=11 | 2
  UOB, NR, BL,n=11 | 1
  UOB, Neg, BL,n=11 | 5
  UOB, 1+, BL,n=11 | 1
  UOB, 2+, BL,n=11 | 0
  UOB, 3+, BL,n=11 | 0
  UOB, Non haemolysed trace, BL,n=11 | 0
  UOB, haemolysed trace, BL,n=11 | 0
  pH, MS, BL, n=11 | 0
  pH, NR, BL, n=11 | 1
  pH, normal result, BL, n=11 | 0
  pH, Neg, BL, n=11 | 0
  pH, 5, BL, n=11 | 2
  pH, 5.5, BL, n=11 | 1
  pH, 6, BL, n=11 | 4
  pH, 6.5, BL, n=11 | 1
  pH, 7, BL, n=11 | 1
  pH, 7.5,BL, n=11 | 1
  pH, 8, BL, n=11 | 0
  pH, 8.5, BL, n=11 | 0
  pH, 9, BL, n=11 | 0
  UP, MS, W24, n=34 | 2
  UP, NR, W24, n=34 | 0
  UP, Neg, W24, n=34 | 32
  UP, Trace, W24, n=34 | 0
  UP, 1+, W24, n=34 | 0
  UP, 2+, W24, n=34 | 0
  UP, 3+, W24, n=34 | 0
  UP, 4+, W24, n=34 | 0
  UG, MS, W24, n=4 | 1
  UG, NR, W24, n=4 | 0
  UG, Neg, W24, n=33 | 29
  UG, normal, W24, n=33 | 3
  UG, 5, W24, n=33 | 0
  UG, 15(1+), W24, n=33 | 0
  UG, 30(2+), W24, n=33 | 0
  UG, 60(3+), W24, n=33 | 0
  UG, 110(4+), W24, n=33 | 0
  UK, MS, W24, n=33 | 1
  UK, NR, W24, n=33 | 0
  UK, Neg, W24, n=33 | 32
  UK, Trace(5), W24, n=33 | 0
  UK, Small(15), W24, n=33 | 0
  UK, Moderate(40), W24, n=33 | 0
  UK, Large(80), W24, n=33 | 0
  UK, Large(160), W24, n=33 | 0
  UOB, MS, W24, n=33 | 1
  UOB, NR, W24, n=33 | 0
  UOB, Neg, W24, n=33 | 31
  UOB, 1+, W24, n=33 | 0
  UOB, 2+, W24, n=33 | 0
  UOB, 3+, W24, n=33 | 0
  UOB, Non haemolysed trace, W24, n=33 | 0
  UOB, haemolysed trace, W24, n=33 | 0
  pH, MS, W24, n=34 | 0
  pH, NR, W24, n=34 | 0
  pH, normal result, W24, n=34 | 0
  pH, Neg, W24, n=34 | 0
  pH, 5, W24, n=34 | 0
  pH, 5.5, W24, n=34 | 4
  pH, 6, W24, n=34 | 10
  pH, 6.5, W24, n=34 | 4
  pH, 7, W24, n=34 | 11
  pH, 7.5,W24, n=34 | 3
  pH, 8, W24, n=34 | 2
  pH, 8.5, W24, n=34 | 0
  pH, 9, W24, n=34 | 0

36. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During Part 1
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect. Medical or scientific judgment should be exercised in other situations.
Time Frame: From Treatment + 1 day up to Week 24 of Part1
Population: Safety Population: all participants who received at least one dose of the investigational product during Part 1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Any AE | 5 | 5 | 5
  Any SAE | 1 | 1 | 0

37. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During Part 2
Description: as for outcome 36
Time Frame: From Treatment + 1 day up to Week 7 of Part 2
Population: Safety Population: all participants who received at least one dose of the investigational product during Part 2 were analyzed.
Measure: Number; unit: Participants
Groups:
- Part 2 (Randomized Period) Cohort 1- Eltrombopag: Participants aged between 12 and 17 years received eltrombopag administered as a tablet for 7 weeks. The starting dose eltrombopag was 37.5 mg QD. The participants of East Asian ancestry began at 12.5 mg QD. The maximum dose allowed was 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
- Part 2 (Randomized Period) Cohort 3- Eltrombopag: Participants aged between 1 to 5 years received eltrombopag administered as a dry powder for oral suspension for 7 weeks. The starting dose of eltrombopag was 1.5 mg/kg QD and the dose calculations were based on the body weight. Participants of East Asian ancestry began at 0.8 mg/kg/day. The maximum dose allowed was 2 mg/kg, as approved by the investigator, and could not exceed 75 mg daily. All participants enrolled in the study underwent individual dose titration based upon platelet response.
Arm/Group | Part 2 (Randomized Period) Cohort 1-Placebo | Part 2 (Randomized Period) Cohort 1- Eltrombopag | Part 2 (Randomized Period) Cohort 2-Placebo | Part 2 (Randomized Period) Cohort 2-Eltrombopag | Part 2 (Randomized Period) Cohort 3-Placebo | Part 2 (Randomized Period) Cohort 3- Eltrombopag
Number analyzed (Participants) | 8 | 16 | 9 | 17 | 4 | 11
Participants
  Any AE | 8 | 13 | 9 | 14 | 3 | 9
  Any SAE | 1 | 1 | 1 | 3 | 0 | 0

38. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During Part 2/3
Description: as for outcome 36
Time Frame: From Treatment + 1 day up to Week 31 of Part2/3
Population: Safety Population: all participants who received at least one dose of the investigational product during Part 2/3 were analyzed
Measure: Number; unit: Participants
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Participants
  Any AE | 22 | 26 | 14
  Any SAE | 3 | 5 | 0

39. Secondary Outcome: Number of Participants With a Change in Visual Acuity and a Change Due to Worsening of Cataracts During Part 1
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. The number of participants with a change in visual acuity and worsening visual acuity due to cataracts since Baseline are presented for Part 1 Follow-up Visits at 3-months (FU3) and at 6-months (FU6). Change in visual acuity since Baseline is displayed under the left eye but applies to both eyes. Change in visual acuity (VA) is categorized as "yes" or "no". Change due to cataracts is categorized as "yes" or "no".
Time Frame: Baseline, 3and 6-mo Follow-up of Part 1
Population: Safety Population: all subjects who have received at least one dose of the investigational product during Part 1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 1 (Dose-Finding Period) Cohort 1 | Part 1 (Dose-Finding Period) Cohort 2 | Part 1 (Dose-Finding Period) Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Change in VA at FU3, no | 1 | 1 | 2
  Change in VA at FU3, yes | 0 | 0 | 1
  Change in VA at FU6, no | 4 | 4 | 5
  Change in VA at FU6, yes | 0 | 0 | 0
  Change due to cataracts at FU3, no | 0 | 0 | 1
  Change due to cataracts at FU3, yes | 0 | 0 | 0
  Change due to cataracts at FU6, no | 0 | 0 | 0
  Change due to cataracts at FU6, yes | 0 | 0 | 0

40. Secondary Outcome: Number of Participants With a Change in Visual Acuity and a Change Due to Worsening of Cataracts
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. Number of participants with a change in visual acuity and change in visual acuity due to the worsening of cataracts since Baseline are presented for Part 2/3 Follow-up Visits at 3-months (FU3) and 6-months (FU6). Change in visual acuity since Baseline is displayed under the left eye but applies to both eyes. Change in visual acuity (VA) is categorized as "yes" or "no". Change due to cataracts is categorized as "yes" or "no".
Time Frame: BL, 3 and 6mo Follow-up of Part 2/3
Population: Safety Population: all subjects who have received at least one dose of the investigational product during Part 2/3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2/3 (Eltrombopag Open-Label Period) Cohort 1 | Part 2/3 (Eltrombopag Open-Label Period) Cohort 2 | Part 2/3 (Eltrombopag Open- Label Period) Cohort 3
Number analyzed (Participants) | 24 | 26 | 15
Participants
  Change in VA at FU3, no | 13 | 17 | 9
  Change in VA at FU3, yes | 4 | 1 | 2
  Change in VA at FU6, no | 16 | 22 | 6
  Change in VA at FU6, yes | 4 | 2 | 3
  Change due to cataracts at FU3, no | 4 | 1 | 2
  Change due to cataracts at FU3, yes | 0 | 0 | 0
  Change due to cataracts at FU6, no | 4 | 2 | 3
  Change due to cataracts at FU6, yes | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs) and serious adverse events (SAEs) are defined as events occuring from the start of the investigational product until the end of treatment (up to Study Week 31)
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who had received at least one dose of the investigational product.
Groups:
- Part 2/ 3 (Eltrombopag Open-Label Period): Par aged between 1 and 17 years (Cohort 1 age group- 12 to 17 years, Cohort 2- 6 to 11 years and Cohort 3-1 to 5 years), completing Part 2 of the study received an Open -Label treatment of eltrombopag administered as a tablet or dry powder for oral suspension in Part 2/3. Par who received eltrombopag during the Randomized Period continued on the same dose unless adjustments were warranted according to the dosing guidelines. Par who received placebo during the Randomized Period followed the starting doses for each age Cohort specified for Part 2.
Arm/Group | Part 1 (Dose-Finding Period) | Part 2 (Randomized Period) -Placebo | Part 2 (Randomized Period) - Eltrombopag | Part 2/ 3 (Eltrombopag Open-Label Period)
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/21 | 4/44 | 8/65
Other Adverse Events (participants affected / at risk) | 15/15 | 20/21 | 36/44 | 62/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose-Finding Period) (N=15) | Part 2 (Randomized Period) -Placebo (N=21) | Part 2 (Randomized Period) - Eltrombopag (N=44) | Part 2/ 3 (Eltrombopag Open-Label Period) (N=65)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Lenticular opacities (Eye disorders) | 0 | 0 | 0 | 1
Vitreous opacities (Eye disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Dose-Finding Period) (N=15) | Part 2 (Randomized Period) -Placebo (N=21) | Part 2 (Randomized Period) - Eltrombopag (N=44) | Part 2/ 3 (Eltrombopag Open-Label Period) (N=65)
Vomiting (Gastrointestinal disorders) | 6 | 6 | 4 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 7 | 17
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3 | 15
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 6
Toothache (Gastrointestinal disorders) | 2 | 0 | 3 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 6 | 15
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 11 | 24
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 8
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 2
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 2
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1 | 3
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infections (Infections and infestations) | 0 | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 3
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal pain (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 9 | 13 | 28
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 5
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 9
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Contusion (Infections and infestations) | 0 | 1 | 1 | 2
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 2 | 4
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Uterine pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 6 | 15
Fatigue (General disorders) | 0 | 2 | 3 | 8
Malaise (General disorders) | 0 | 0 | 1 | 2
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 2
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 2
Local swelling (General disorders) | 0 | 0 | 0 | 2
Feeling jittery (General disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 1
Tic (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Haematotympanum (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Decreased appetite (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 4
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.